

## ISTITUTO DI RICERCHE FARMACOLOGICHE "MARIO NEGRI" IRCCS

Study Name BAROCCO

SAP

version 1.0 - 11 December 2017

### STATISTICAL ANALYSIS PLAN

**STUDY NAME: BAROCCO** 

TRIAL CODE: IRFMN-OVA3-7289

EudraCT: 2016-003964-38

**Best Approach in Resistant-Ovarian-Cancer with-Cediranib-Olaparib:** an Italian multicenter randomized phase II study of weekly paclitaxel vs. Cediranib-Olaparib with continuous schedule vs. Cediranib-Olaparib with intermittent schedule in patients with platinum resistant high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer.

Study Sponsor:

Study Statistician:

Mario Negri Gynecologic Oncology

Group - MaNGO

IRCCS – Istituto di Ricerche farmacologiche Mario Negri

Via La Masa, 19 - 20156 Milano (Italy)

Alvisi Maria Francesca, MSc.

Laboratory of methodology for clinical

research

Department of Oncology

IRCCS Istituto di Ricerche farmacologiche

Mario Negri

Via La Masa, 19 - 20156 Milano (Italy)

DOCUMENT: Statistical Analysis Plan

STUDY: BAROCCO
DOCUMENT VERSION: 01
DATE: 11/12/2017

AUTHOR: Maria Francesca Alvisi

# **Version History**

This version of the *Statistical Analysis Plan* becomes effective on the date of final approval. If changes are made that affect the document's content or approach, a revised, complete document must be issued for re-approval by the roles of the approvers of the original document or their designated representatives. A description of those changes with revision number is noted in the revision log below:

| Version | Date | Reason for<br>issue/change | Author | Signature |
|---|---|---|---|---|
| 01 | 11/12/2017 | Initial Document | Maria Francesca Alvisi | Mode Francisco Alina |

| Version | Date | Reason for issue/change | Reviewer | Signature |
|---------|------|-------------------------|----------|-----------|
| 01 | | Initial Document | | |

| Version | Date | Reason for<br>issue/change | Approvers | Signature |
|---------|------|----------------------------|-----------|-----------|
| 01 | | Initial Document | | |

### LIST OF ABBREVIATIONS

95%CI 95% confidence interval

CR Complete Response

CSR Clinical study report

e-CRF Electronic- case record form

FACT-O Functional Assessment of Cancer Therapy-Ovarian

HR Hazard ratio

ICH International Conference on Harmonization

ITT Intent-to-treat

ORR Overall response rate

OS Overall survival

PFS Progression free survival

PD Progression of Disease

PP Per-ptotocol

PR Partial Response

PRO Patient reported outcome

RECIST Response Evaluation Criteria in Solid Tumours

SADR Safety Adverse Drug Reaction

SAE Serious Adverse Event

SD Stable Disease

SE Safety evaluable

SOC System organ class

SUSAR Suspected Unexpected Serious Adverse Reaction

WHO World health organization

### **TABLE OF CONTENTS PAGE** VERSION \_\_\_\_\_\_2 INTRODUCTION......6 1. GENERAL DESCRIPTION OF FINAL STUDY REPORT......6 2. 2.1 Responsibilities......6 2.2 Structure 6 2.3 Text .......7 2.3.1 2.3.2 SAS Outputs......7 3. STUDY OBJECTIVES......9 Efficacy objectives.....9 Primary objective.....9 Secondary objective ......9 3.1.2 Safety objectives ......9 3.2 Compliance endpoints......10 3.3 4. INVESTIGATIONAL PLAN......10 4.1 4.2 4.1 Interim Analysis......12 5. DATA SUMMARIES AND STATISTICAL ANALYSIS......13 5.1 Trial closure and data cut-off......13 5.1.1 5.1.3 General Considerations......13 5.1.4 Methods for Handling Withdrawals, Missing Data and Outliers......14 5.2 5.3 5.4 Disposition of Subjects ......17 Inclusion and Exclusion Criteria......18 5.4.2 5.4.3 5.5 Data Sets Analyzed ......18

| Statistical | Analysis | Plan |
|-------------|----------|------|

| - | 70.0 | 000 |
|---|------|-----|

| 200 | |
|---|---|
| 5.5.3 Measurement of Treatment Compliance | 19 |
| · | |
| 5.5.4.2 Objective Response Rate | 20 |
| 5.5.4.5 Quality of Life | 21 |
| 5.6.1 Number of evacuations per day | 22 |
| · · | |
| APPENDIX A: TABLES OF SECTION 14 OF THE CSR | 25 |
| APPENDIX B: LISTINGS OF SECTION 16.2 OF THE CSR | 85 |
| APPENDIX C: FIGURES TEMPLATE | 107 |
| | 5.5.3 Measurement of Treatment Compliance |

### 1. INTRODUCTION

This document outlines the statistical methods for the analysis of data collected under Protocol No. IRFMN-OVA3-7289 and based on Version 1 of the Final Protocol dated 20/11/2017 and on the Final Version of the electronic- case record form (e-CRF) dated 11/10/2016.

The main objective of this document is to provide guidance for the production of the Clinical Study Report (CSR), including post-text tables, post-text listings (related to specific tables) and other listings (for all patients and all variables included in the Clinical Data Base).

### 2. GENERAL DESCRIPTION OF FINAL STUDY REPORT

The CSR of BAROCCO will fulfill all recommendations given in the guideline ICH topic E3 "Note for Guidance on Structure and Content of Clinical Study Report" (CPMP/ICH/137/95).

American English will be used for writing the CSR.

The core of the CSR will be written with Microsoft Word version 2016; all data summaries (tables) and listings will be prepared by using SAS Version 9.4.

The choice of the population(s) included in the table will depend on the considered variable.

### 2.1 Responsibilities

The CSR of the present study will be written by the statistician of the study. The structure of the CSR (see section 2.2 of this document) will be according to the guideline ICH topic E3.

### 2.2 Structure

The CSR will be divided in sections, titled and numbered as requested by the above mentioned guideline. The most relevant sections concerning study results are illustrated below.

| Topics | Section |
|-----------------------------------------------|---------------|
| Disposition of Patients | 10.1 |
| Protocol Deviations | 10.2 |
| Data Sets Analyzed | 11.1 |
| Demographics & Other Baseline Characteristics | 11.2 |
| Measurements of Treatment Compliance | 11.3 |
| Efficacy Results | 11.4 |
| Adverse Events | 12.2 |
| Post-text Tables and Listings | 14 |
| Patient Data Listings | Appendix 16.2 |

## 2.3 Format

### 2.3.1 Text

All the pages of the CSR core (text) should contain the following information:

- Protocol identification;
- Page number;
- Specification of document version and date;

## 2.3.2 SAS Outputs

All tables and listings of the CSR will be generated by SAS version 9.4.

When not otherwise specified (in the SAS outputs), location indicators, percentages and standard deviations (SDs) will be rounded to the first decimal digit.

Dates will always be displayed as ddmmyyyy.

## Format of SAS Outputs

Statistical Analysis Plan

**BAROCCO** 

As for the format of the SAS outputs (tables and listings), all the pages should contain the following information:

- Protocol identification;
- Specification of document version;
- Page number;
- Date when the output was generated;

# Table/Listing Numbering and Naming of corresponding SAS programs

Patients Data Listings (for all patients and all variables included in the data base) will be included in Appendix 16.2 of the CSR.

Listings of all the individual patient data collected during the study will be included in Appendix 16.2 of the CSR (more details are given in Appendix 2 of this document).

Listings will be numbered as follows:

<Section>.<Listing Number>, where:

- <Section> is the number identifying the CSR section referencing the listing;
- o <Listing number> indicates the sequence of the listings in each section.

The SAS program generating these listings will be named as

AL. < Section > . < Listing number > . sas, and the corresponding output as

AL. <Section>. <Listing number>.rtf, where

- AL= Appendix Listings;
- <Section> is the number identifying the CSR section referencing the listing;
- o <Listing number> is the number indicating the listing sequence.

### 3. STUDY OBJECTIVES

This section is a draft of Section 8 of the CSR (see guideline ICH topic E3).

## 3.1 Efficacy objectives

## 3.1.1 Primary objective

The study primary objective is to compare the efficacy of Olaparib and Cediranib vs. weekly paclitaxel in terms of progression free survival (PFS) in platinum refractory or resistant recurrent ovarian cancer.

PFS is defined as the time from randomization to the date of first progression or death for any cause, whichever comes first.

Progression will be established as the objective radiological disease progression according to RECIST 1.1 or to clinical assessment.

# 3.1.2 Secondary objective

- Objective Response Rate (ORR), defined as the percentage of patients with an objective response as determined by RECIST 1.1
- PFS2 defined as time from randomization to second disease progression according to RECIST 1.1 or to clinical assessment, or death by any cause.
- Overall Survival (OS), defined for each patient as the time from randomization to the date of death for any cause.
- Quality of Life evaluated by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) questionnaire.

### 3.2 Safety objectives

The primary objective for safety is to compare the safety of Olaparib and Cediranib as intermittent vs. continuous regimen in terms of number of evacuations per day.

Secondary objectives are:

 Maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 4.0; Statistical Analysis Plan BAROCCO

- patients experiencing grade 3-4 toxicities for each toxicity;
- type, frequency and nature of SAEs;
- patients with at least a SAE;
- patients with at least a SADR;
- patients with at least a SUSAR.

## 3.3 Compliance endpoints

Compliance will be evaluated in terms of number of:

- administered cycles;
- · reasons for discontinuation and treatment modification;
- dose intensity.

### 4. INVESTIGATIONAL PLAN

This section is a draft of Section 9 of the CSR (see guideline ICH topic E3). For further details refer to the study protocol.

### 4.1 General trial design

This is a Phase II, randomized, multi-center study with two experimental arms, Cediranib-Olaparib with continuous schedule and Cediranib-Olaparib with intermittent schedule. Weekly paclitaxel is the comparator arm, due to its known efficacy in platinum resistant/refractory disease.

All patients not previously tested for the presence of BRCA1-2 germline mutations will undergo BRCA test. However, both mutated and not mutated women will be included in the study protocol.

Randomization will use a biased-coin minimization procedure having as stratification factors BRCA1-2 genes status (mutated vs. wild-type vs. still unknown), prior chemotherapy (1-2 vs.  $\geq$  3 lines) and previous treatment with antiangiogenic drugs (yes vs. no). Patients will be randomized in a 1:1:1 ratio to the treatments as specified below:

ARM A: Paclitaxel 80 mg/mq every week.

**ARM B:** Cediranib 20 mg/day + Olaparib 600 mg / day (i.e. 300 mg BD) given every day.

**ARM C:** Cediranib 20 mg/day given 5 days per weeks + Olaparib 600 mg / day (i.e. 300 mg BD) given 7 days per weeks.

Figure 1. Study flow-chart



\*For Arm A (weekly Paclitaxel): maximum 24 weeks.

BD:twice daily

Progression will be established as the radiological disease progression according to RECIST 1.1 or as clinical progression in case radiological evaluation is not feasible due to clinical condition.

All patients should have RECIST assessments until documented evidence of radiological progression in accordance with RECIST 1.1, irrespective of treatment decisions (i.e. RECIST follow up until progression even if a patient discontinues study treatment prior to progression and/or receives a subsequent therapy prior to progression).

Disease assessments will be scheduled every 8 weeks (+/-1 week) from randomization for all treatment duration and every 12 weeks (+/-1 week) thereafter.

# 4.2 Sample size determination

Assuming a median PFS in the control arm of 3.4 months (AURELIA trial control group), this study is designed to detect a HR of 0.51 that corresponds to an advantage in PFS median of 3.3 months. With one-sided 5% significance level and with at least 80% power, approximately 60 patients (55 events) for each comparison are estimated to be enrolled. Considering the two pre-planned comparisons (intermittent schedule vs Paclitaxel and continuous schedule vs Paclitaxel) a total of 90 eligible patients are needed. Taking into account a 10% of patients not evaluable for the primary endpoint, it will be necessary to enroll approximately 100 patients.

# 4.1 Interim Analysis

There are no formal interim analyses planned for this study.

### 5. DATA SUMMARIES AND STATISTICAL ANALYSIS

The following section is a draft of Sections 10.1 (Disposition of Patients), 10.2 (Protocol Deviations), 11 (Efficacy evaluation – see detailed sub-sections in paragraph 5.5 of the present document) and 12 (Safety evaluation – see detailed sub-sections in paragraph 5.6 of the present document) of the CSR (see also guideline ICH topic E3).

### 5.1 Definitions and conventions

### 5.1.1 Trial closure and data cut-off

The final analysis will be performed after reaching the PFS target number of events and after cleaning data in order to preserve the accurate frozen database.

#### 5.1.2 Protocol violations and deviations

Major violations in the eligibility criteria, minor deviation and study conduction will be evaluated on a case by case basis in a pre-analysis meeting considering the following points:

- 1. Unfulfilled inclusion criteria
- 2. Subject enrollment and/or treatment in the presence of Exclusion Criteria
- 3. Treatment with unauthorized concomitant medication
- 4. Treatment regimen violations.

### 5.1.3 General Considerations

- Continuous variables will be described including number of observations, mean, standard deviation (SD), median, ranges (minimum and maximum) and number of missing values;
- Categorical variables will be described including the frequency and percentage of subjects in each category. In general, the denominator for

the percentage calculation should be the total number of subjects in the relevant analysis set, unless otherwise specified. Percentages are to be rounded to one decimal place;

- Response will be provided as the absolute and relative frequencies of patients with CR, PR, SD and PD according to RECIST. 95% CIs of response rate will be computed by means of exact binomial methods.
- Time-to-event variables (PFS, OS, PFS2) will be described with the Kaplan-Meier method. KM estimates for median and quartile event times, and event-free rates at selected times will be calculated. Cox regression model will be performed in order to evaluate the reduction of the risk in the differences in PFS, PFS2 and OS between arms, by including stratification variables and other clinical-biological features as covariates. Results will be presented as hazard ratios (HRs) and their 95% confidence intervals (95% CIs) unless otherwise specified.

# 5.1.4 Methods for Handling Withdrawals, Missing Data and Outliers

Missing values will be defined as not imputed, unless otherwise specified.

For time to event analysis calculate incomplete or missing dates of disease progression or death using the following approach:

- if the month and the year are reported, assign the 15th day of the month by default;
- if the entire date is unknown, assign the day following the last information available, in which the subject was known to be progression free or alive.

### 5.2 Analysis sets

The analysis sets described below will be considered for the analysis, as follows:

<u>All Subjects Analysis Set:</u> the All Subjects Analysis Set is defined as all participants who provided informed consent and were enrolled in the study. The listings of all variables will be based on the All Subjects Analysis Set.

**Intent-to-Treat (ITT) Analysis Set:** the ITT analysis set is defined as all randomized patients, without major violations of eligibility criteria. Patients will be analyzed according to randomization arm.

Major violations in the eligibility criteria will be evaluated on a case by case basis in a pre-analysis meeting in order to define the population.

**Per-protocol (PP) Analysis Set:** the PP analysis set is defined as all patients of the ITT analysis set, who received at least 4 weeks of treatment, unless they interrupted before for disease progression or death. Patients randomized to the control arm, receiving the experimental treatment and patients randomized to the experimental arm, receiving the control treatment will be excluded.

<u>Safety 1 Analysis Set:</u> the Safety 1 Analysis Set is defined as all patients included of the ITT Analysis Set, who were randomized to the two experimental arms, excluding patients who interrupted before 4 weeks, unless the interruption is due to diatrrhea. Patients randomized to the continue schedule (arm B), receiving the intermittent schedule (as arm C) and patients randomized to the intermittent schedule, receiving the continue schedule will be excluded.

<u>Safety 2 Analysis Set:</u> the Safety 2 Analysis Set is defined as all patients included of the ITT Analysis Set, who received at least one dose of study treatment, whether withdrawn prematurely or not. Patients will be considered in the treatment arm they actually received.

**Overall Response Rate (ORR) Analysis Set:** the ORR analysis set is defined as all patients included in the ITT analysis set, receiving at least one dose of study treatment and with at least one radiological assessment. Radiological assessment will be evaluated in accordance to RECIST criteria.

**Compliance analysis set:** the Compliance Analysis Set included all subjects of ITT analysis. Patients will be considered in the treatment arm they actually received. The Compliance Analysis Set is used for the compliance analyses.

<u>Patient reported outcome (PRO) Analysis Set:</u> the PRO Analysis Set includes all subjects of ITT analysis set with the evaluation of FACT-O questionaires.

# 5.3 **Study-Population and Strata to be used**

Tables will be created by strata (column) and applied to specific study population (patients/records contributing to table) according to the criteria described in the table below.

Table - Analysis sets and Strata to be applied

| SECTION | TABLES | ANALYSIS<br>SET | STRATA |
|---|---|---|---|
| ENROLMENT AND DISPOSITION OF PATIENTS | 14.1.1.x | ALL RANDOMIZED PATIENTS | TREATMENT ARM |
| DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 14.1.2.x | ITT | TREATMENT ARM |
| MEASUREMENT OF TREATMENT COMPLIANCE | 14.2.1.x | COMPLIANCE | TREATMENT ARM |
| EFFICACY | | | TREATMENT ARM |
| Progression Free Survival | 14.2.2.x | ITT AND PP | |
| Objective Response Rate | 14.2.3.x | ORR | |
| Second Progression Free Survival | 14.2.4.x | ITT AND PP | |
| Overall Survival | 14.2.5.x | ITT AND PP | |
| Quality of Life | 14.2.6.x | PRO | |
| SAFETY | | | |
| Primary Safety analyses | 14.3.1.1 | SAFETY 1 | TREATMENT ARM |
| (intermittent vs. continuous) | | | (B vs. C) |
| Secondary Safety analyses | 14.3.1.x | SAFETY 2 | TREATMENT ARM |

# 5.4 Enrollment and Disposition of Patients

# **5.4.1** Disposition of Subjects

A summary table will be provided showing the number of randomized patients, the number of withdrawn and the reasons for withdrawal for the overall population, grouped by study treatment.

Subject disposition will be described using the All Subjects Analysis Set.

Subject disposition is summarized in Appendix A, Table 1 and listed by subject in Appendix B, Listing 1.

### 5.4.2 Inclusion and Exclusion Criteria

Inclusion and exclusion criteria will be described using the *All Subjects Analysis Set*.

Inclusion and exclusion criteria is listed by subject in Appendix B, *Listing 3* and *Listing 4*.

### 5.4.3 Protocol Violations and Deviations

A summary table will be provided showing the number and type of minor and major deviations for the overall population, grouped by study treatment.

Protocol deviations will be described using the All Subjects Analysis Set.

Protocol deviations are summarized in Appendix A, *Table 2* and listed by subject in Appendix B, *Listing 2*.

# 5.5 Efficacy evaluation

### 5.5.1 Data Sets Analyzed

Two summary tables will be provided showing:

- The total number of patients included in each analysis set for the overall population, grouped by study treatment.
- The number of patients by center included in each analysis set for the overall population, grouped by study treatment.

Data sets analyzed are summarized in Appendix A, Table 3 and Table 4.

# 5.5.2 Demographics and other baseline characteristics

A summary table will be provided showing demographics and other patients' baseline characteristics for the overall population, grouped by study treatment.

Demographics and other patients' baseline characteristics will be described using the *ITT analysis set*.

Demographic and other baseline characteristics are summarized in Appendix A, *Table 5* and listed by subject in Appendix B, *Listing 6*.

A summary table will be provided showing tumor characteristics for the overall population, grouped by study treatment.

Tumor characteristics will be described using the *ITT analysis set*.

Tumor characteristics are summarized in Appendix A, *Table 6* and listed by subject in Appendix B, *Listing 7*.

A summary table will be provided showing previous therapies for the overall population, grouped by study treatment.

Previous therapies will be described using the *ITT analysis set*.

Previous therapies are summarized in Appendix A, *Table 7* and *Table 8* listed by subject in Appendix B, Listing 8.

### **5.5.3 Measurement of Treatment Compliance**

Summary tables will be provided for the overall population and grouped by study treatment showing:

- the number of patients who never started or discontinued treatment
- the reasons for not starting the treatment
- the reasons for treatment interruption

- the number of completed cycles in subjects who discontinued treatment
- the dose intensity: which is defined as, for each agent separately, percent of dose received related to expected dose as following:

$$dose\ intensity = \frac{total\ dose\ received\ in\ mg/m^2}{expected\ dose\ in\ mg/m^2\times total\ number\ of\ expected\ cycles}$$

Treatment compliance will be described using the Compliance analysis set.

Treatment compliance is summarized in Appendix A, *Table 9*, *Table 10*, *Table 11* and listed by subject in Appendix B, *Listing 9* and *Listing 10*.

### 5.5.4 Efficacy Results

## 5.5.4.1 Progression Free Survival

PFS will be analyzed using the *ITT Analysis Set* first, and as secondary analyses, PFS will be analysed on *PP Analysis Set*.

PFS is summarized in Appendix A, Table 12 and .

Cox Models (univariate and multivariate analysis) are presented in Appendix A, *Table 14* and *Table 15*.

Kaplan-Meier curves are presented in Appendix C, Figure 2 and Figure 3. Efficacy data is listed by subject in Appendix B, Listing 11.

# 5.5.4.2 Objective Response Rate

ORR will be analyzed using ORR Analysis Set.

ORR is summarized in Appendix A, Table 16 and Table 17.

Efficacy data is listed by subject in Appendix B, Listing 13.

# 5.5.4.3 Second Progression Free Survival

PFS2 will be analyzed using the *ITT Analysis Set* first, and as secondary analyses, PFS2 will be analysed on *PP Analysis Set*.

PFS2 is summarized in Appendix A, Table 18 and Table 19.

Cox Models (univariate and multivariate analysis) are presented in Appendix A, *Table 20* and *Table 21*.

Kaplan-Meier curves are presented in Appendix C, *Figure 4* and *Figure 5*. Efficacy data is listed by subject in Appendix B, *Listing 12*.

### 5.5.4.4 Overall Survival

OS will be analyzed using the *ITT Analysis Set* first, and as secondary analyses, OS will be analysed on *PP Analysis Set*.

OS is summarized in Appendix A, Table 22, Table 23.

Cox Models (univariate and multivariate analysis) are presented in Appendix A, Table 24 and Table 25.

Kaplan-Meier curves are presented in Appendix C, *Figure 6 and Figure 7*. Efficacy data is listed by subject in Appendix B, *Listing 11*.

### 5.5.4.5 Quality of Life

Quality of Life evaluated by the Functional Assessment of Cancer Therapy-Ovarian (FACT-O) questionnaire. Change scores in quality of life (i.e. differences from baseline to each visit) will be calculated and described at every visit and at the time of study discontinuation, for each domain and within each arm.

A mixed model will be performed in order to assess differences in quality of life scores among groups and the interaction between time and treatment.

PRO will be analyzed using the PRO Analysis Set.

FACT-O scores are summarized for four evaluation in *Table 26*: baseline (T0), after 4 weeks (T1), after 8 weeks (T2) and after 12 weeks (T3).

Changes from baseline are presented in *Table 27* and mixed models are reported in *Table 28*. PRO data is listed by subject in Appendix B, *Listing 15* and *Listing 16*. The scores for each subscale will be calculated according the scoring system of FACT-O.

# 5.6 Safety Evaluation

The primary endpoint for safety is the number of evacuations per day.

Secondary endpoints of safety are:

- the maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 4.0;
- the number of patients experiencing grade 3-4 toxicity for each toxicity;
- type, frequency and nature of SAEs;
- patients with at least a SAE; patients with at least a SADR;
- patients with at least a SUSAR.

Adverse Events (AEs) will be coded using the MedDRA coding dictionary and graded using the NCI-CTCAE scale, version 4.0

The chi-squared test for trend will be used to compare the maximum grade for each type of adverse event by treatment arm.

The primary safety analyses will be done using the Safety 1 Analyses set.

The secondary analyses will be conducted using the Safety 2 Analysis set.

### 5.6.1 Number of evacuations per day

The number of evacuations per day analysis will be conducted on the *Safety* 1 analysis set excluding patients who interrupted the treatment before 4 weeks, unless the interruption is due to diarrhea.

In case both arms will demonstrate the superiority over control arm in terms of PFS, the best schedule will be selected based on safety profile considering in particular the mean number of evacuations per day. The difference on mean number of evacuations per day will be tested through a t-test test for two independent groups. If the normality assumptions cannot be assumed a non-parametrical test will be performed.

The mean number of evacuations per day will be presented in Appendix A, *Table 29*. Changes on mean number of evacuations per day will be presented in Appendix A, *Table 30* and Appendix B, *Listing 17*.

For each patient and for each type of adverse event, the worst degree ever suffered during treatment will be used for the analysis.

### 5.6.2 Treatment Tolerability

The maximum grades of each adverse event per subject will be used to analyze treatment tolerability.

Adverse events related to the study drugs according to the investigators judgment are summarized in Appendix A, *Table 31*. MedDRA terms will be used.

Treatment tolerability data is listed by subject in Appendix B, *Listing 18* and *Listing 19*.

### **5.6.3 Serious Adverse Events**

The assessment of safety will be mainly based on adverse reactions (ARs) and the frequency and nature of SAEs and will be conducted on the Safety 2 Analysis Set.

SAEs will be summarized by presenting the number and percentage of patients having any SAE and having an SAE in each system organ class. Other information collected (e.g. severity or suspected relationship to study medication) will be listed as appropriate.

A summary table will be provided showing SAEs occurred during the study for the overall population, grouped by study treatment.

SAEs occurred during the study are summarized in Appendix A, Table 32, Table 33, Table 34, Table 35 and Table 36.

All SAEs will be listed by subject in Appendix B, Listing 20 .

# 6. APPENDIX A: TABLES OF SECTION 14 OF THE CSR

Overall content of Section 14 of the CSR (see guideline ICH topic E3):

- 14.1 Demographic Data
- 14.2 Efficacy Data
- 14.3 Safety Data
- 14.3.1 Displays of Adverse Events
- 14.3.2 Listings of Deaths, Other Serious and Significant Adverse Events
- 14.3.3 Narratives of Deaths, Other Serious and Significant Events

| Table<br>Number | Table Title | Section of the CSR | Page |
|---|---|---|---|
| Table 1 | Subjects Disposition – All Subjects Analysis Set (table 14.1.1.1 CSR) | 14.1 | 28 |
| Table 2 | Protocol Violations and Deviations – All Subjects Analysis Set (table 14.1.1.2 CSR) | 14.1 | 29 |
| Table 3 | Data Analysis Sets - All Subjects<br>Analysis Set (table 14.1.1.3 CSR) | 14.1 | 29 |
| Table 4 | Recruitment, Analysis set and Allocation to treatment per Study Centre (table 14.1.1.4 CSR) | 14.1 | 31 |
| Table 5 | Demographic and Baseline<br>Characteristics – ITT Analysis Set (table<br>14.1.2.1 CSR) | 14.1 | 32 |
| Table 6 | Tumour Characteristics – ITT Analysis<br>Set (table 14.1.2.2 CSR) | 14.1 | 35 |
| Table 7 | Previous therapies – ITT Analysis Set (table 14.1.2.3 CSR) | 14.1 | 37 |
| Table 8 | Previous therapies – Last Platinum free interval – ITT Analysis Set (table 14.1.2.4 CSR) | 14.1 | 41 |
| Table 9 | Treatment Compliance – ITT Analysis Set (table 14.2.1.1 CSR) | 14.2 | 42 |
| Table 10 | Number of completed cycles in subjects who have discontinued the treatment – Compliance Analysis Set (table 14.2.1.2 CSR) | 14.2 | 44 |
| Table 11 | Dose intensity – Compliance Analysis Set (table 14.2.1.3 CSR) | 14.2 | 45 |
| Table 12 | Progression Free Survival – ITT Analysis<br>Set (table 14.2.2.1 CSR) | 14.2 | 47 |

| Table | Table Title | Section | D |
|---|---|---|---|
| Number | Table Title | of the<br>CSR | Page |
| Error!<br>Reference<br>source not<br>found. | | 14.2 | Error!<br>Bookmark<br>not<br>defined. |
| Table 14 | Progression Free Survival – Cox models – ITT Analysis Set (table 14.2.2.3 CSR) | 14.2 | 51 |
| Table 15 | Progression Free Survival – Cox models – PP Analysis Set (table 14.2.2.4 CSR) | 14.2 | 52 |
| Table 16 | Response to treatment – ORR Analysis<br>Set <i>(table 14.2.3.1 CSR)</i> | 14.2 | 53 |
| Table 17 | Objective response rate – ORR Analysis<br>Set <i>(table 14.2.3.2 CSR)</i> | 14.2 | 54 |
| Table 18 | Second Progression Free Survival – ITT<br>Analysis Set (table 14.2.4.1 CSR) | 14.2 | 55 |
| Table 19 | Second Progression Free Survival – PP<br>Analysis Set <i>(table 14.2.4.2 CSR)</i> | 14.2 | 56 |
| Table 20 | Second Progression Free Survival – Cox models - ITT Analysis Set (table 14.2.4.3 CSR) | 14.2 | 57 |
| Table 21 | Second Progression Free Survival – Cox models - PP Analysis Set (table 14.2.4.4 CSR) | 14.2 | 58 |
| Table 22 | Overall Survival – ITT Analysis Set (table 14.2.5.1 CSR) | 14.2 | 59 |
| Table 23 | Overall Survival – PP Analysis Set <i>(table 14.2.5.2 CSR)</i> | 14.2 | 60 |
| Table 24 | Overall Survival – Cox models - ITT<br>Analysis Set <i>(table 14.2.5.3 CSR)</i> | 14.2 | 60 |
| Table 25 | Overall Survival – Cox models - PP<br>Analysis Set <i>(table 14.2.5.4 CSR)</i> | 14.2 | 62 |
| Table 26 | Quality of life - PRO Analysis Set (table 14.2.6.1 CSR) | 14.2 | 63 |
| Table 27 | Quality of life - Change from baseline - PRO Analysis Set (table 14.2.6.2 CSR) | 14.2 | 66 |
| Table 28 | Quality of life – Mixed model for differences from baseline - PRO Analysis Set (table 14.2.6.3 CSR) | 14.2 | 70 |
| Table 29 | Number of evacuations per day – Safety<br>1 Analysis Set (table 14.3.1.1 CSR) | 14.3 | 71 |
| Table 30 | Change of evacuations per day – Safety<br>1 Analysis Set (table 14.3.1.2 CSR) | 14.3 | 75 |
| Table 31 | Adverse reactions – Safety 2 Analysis<br>Set (table 14.3.1.3 CSR) | 14.3 | 76 |

| Table<br>Number | Table Title | Section<br>of the<br>CSR | Page |
|---|---|---|---|
| Table 32 | Overview of Serious Adverse Events –<br>Safety 2 Analysis Set (table 14.3.1.4<br>CSR) | 14.3 | 78 |
| Table 33 | Description of Serious Adverse Events (SAEs) – Safety 2 Analysis Set (table 14.3.1.5 CSR) | 14.3 | 79 |
| Table 34 | Description of Serious Adverse Events (SAEs) by MedDRA – Safety 2 Analysis Set (table 14.3.1.6 CSR) | 14.3 | 80 |
| Table 35 | Description of Serious Adverse Drug<br>Reactions (SADRs) - Safety 2 Analysis<br>Set (table 14.3.1.7 CSR) | 14.3 | 82 |
| Table 36 | Description of Serious Adverse Drug<br>Reactions (SADRs) by MEdDra – Safety 2<br>Analysis Set (table 14.3.1.8 CSR) | 14.3 | 84 |

Statistical Analysis Plan

BAROCCO

Table 1. Subjects Disposition - All Subjects Analysis Set (table 14.1.1.1 CSR)

| | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | (%) N | (%) N | (%) N | (%) N |
| Patients discontinued | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Main reason for discontinuation: | | | | |
| Disease Progression | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Toxicity | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Death | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Subject refusal | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Medical decision | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Major violation | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Lost to follow-up | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Other | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |

**Legend:** ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects.

Statistical Analysis Plan BAROCCO

Overall N=XX  $\stackrel{>}{\sim}$   $\stackrel{>}{\sim}$   $\stackrel{>}{\sim}$ × Table 2. Protocol Violations and Deviations – All Subjects Analysis Set (table 14.1.1.2 CSR) ARM C X=Z × × × ×  $\stackrel{\times}{\sim}$ ARM B XXII × ×  $\stackrel{\times}{\times}$ × × **ARM A** XX=N ×  $\stackrel{>}{\sim}$  $\stackrel{\times}{\sim}$ X × Any protocol violation such to exclude the subject from Description of 3 minor protocol violation / deviation Description of 2 minor protocol violation / deviation Description of 1 minor protocol violation / deviation Description of 4 minor protocol violation / deviation Violations of the eligibility criteria Any minor protocol deviation: Number of patients any analysis set: Subject status

Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects

BAROCCO

Table 3. Data Analysis Sets - All Subjects Analysis Set (table 14,1.1.3 CSR)

| | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | N=XX | N=XX | XX=N | N=XX |
| All subjects analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | (x.xx) XX |
| Intent-to-treat analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Per Protocol analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Safety 1 analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Safety 2 analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Overall Response Rate analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Compliance analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Patients reported outcome analysis set - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |

Recruitment, Analysis set and Allocation to treatment per Study Centre (table 14.1.1.4 CSR) Table 4.

| Table 4. | 4 | | Recruitment, Analysis set an | ţIJ | ent, | An | alX | SIS | Set | and | 4 | SCO | 101 | טיר | d Allocation to treatment | | en: | e<br>C | ה<br>ה | | ۲ | per study centre (GDIE 14.1.1.4 | 2 | 906 | 14 | 7.7 | | 35 | | | İ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Cen | A | Sub | Subjects<br>set | | H | ITT S | set | | <b></b> | PP se | et | ~• | Safety | + | set | S | Safety | y 2 set | ë | U | omi | Compliance<br>set | e<br>O | | ORR | set | | | PRO | set | |
| _ | 4 =<br>4 × 4 | A Z A | AR M | A E O | A =<br>A Σ A | A A A A B A | | A E O | A A A A | A A R | A = Ω | <b>∀</b> = | AΣΑ | AR<br>B | A E O | ⋖= | A Z A | AR<br>M | ARΩ | <b>V</b> = | A Z A | AR<br>B | AR C | <b>A</b> = | A Z A | A Σ a | A Z O | <b>V</b> = | ARA | A Z a | AΣΩ |
| Cen<br>tre<br>1 | ×× | × | × | ×× | ×× | | × | | ×× | × | × | ×× | × | × | × | ×× | × | × | × | ×× | × | × | × | ×× | × | × | × | ×× | × | × | × |
| Cen<br>tre<br>2 | ×× | × | × | ×× | ×× | × | × | ××<br>× | × | × | × | ×× | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × |
| Cen<br>tre<br>3 | ×× | × | × | ×× | ×× | × | × | | ×× | × | × | ×× | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × |
| Cen<br>tre<br>4 | × | × | × | × | ×× | × | × | ××<br>× | × | × | × | ×× | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | ҳ | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × |
| Cen<br>tre<br>5 | ×× | × | × | × | ×× | × | × | | ×× | × | × | ×,× | × | × | × | $\times \times$ | × | × | × | $\times \times$ | ҳ | × | × | ×× | × | × | × | ×× | × | × | × |
| Cen<br>tre<br>6 | × | × | × | × | ×× | × | | ×× | ×× | × | ×× | ×× | × | × | × | ×× | × | × | × | $\times \times$ | × | × | × | $\times \times$ | × | × | × | ×× | × | × | × |

Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; n: number of subjects

Table 5. Demographic and Baseline Characteristics – ITT Analysis Set (table 14.1.2.1 CSR)

| Number of patients - n (%) | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Age | | | | |
| Mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X -<br>XX-X) | XX.X (XX.X<br>- XX-X) |
| Min – max | XX.X -<br>XX.X | xx.x - xx.x | XX.X - XX.X | XX.X<br>XX.X |
| Missing | xx | xx | xx | xx |
| Performance status – n (%) | | | | |
| 0 | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| 1 | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| Missing | xx | xx | xx | XX |
| Weight (Kg) | | | | |
| Mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X -<br>XX-X) | XX.X (XX.X<br>- XX-X) |
| Min – max | XX.X -<br>XX.X | xx.x - xx.x | XX.X - XX.X | XX.X –<br>XX.X |
| Missing | xx | xx | xx | xx |
| Height (cm) | | | | |
| Mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X -<br>XX-X) | XX.X (XX.X<br>- XX-X) |
| Min – max | XX.X -<br>XX.X | xx.x - xx.x | XX.X - XX.X | XX.X –<br>XX.X |
| Missing | XX | XX | xx | xx |
| Race - n (%) | | | | |
| Caucasian | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| Black | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| Asian | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| Other | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| Missing | XX (XX) | XX (XX) | XX (XX) | XX (XX) |
| BRCA 1 mutational status - n (%) | | | | |
| Mutated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Wild-type | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

| Number of patients - n (%) | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Unknown | xx | XX | XX | xx |
| Missing | xx | xx | xx | xx |
| BRCA 2 mutational status - n (%) | | | | |
| Mutated | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Wild-type | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | xx | XX | XX | xx |
| Missing | xx | XX | xx | xx |
| CA-125 (U/mL) | | | | |
| Mean (SD) | XX.X<br>(XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X<br>- XX-X) | XX.X (XX.X -<br>XX-X) | XX.X (XX.X<br>- XX-X) |
| Min - Max | XX.X<br>XX.X | xx.x - xx.x | xx.x - xx.x | XX.X -<br>XX.X |
| Missing | XX | XX | XX | xx |
| Relevant disease - n (%) | | | | |
| No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX | xx | XX | xx |
| Start of disease - n (%) | | | | |
| Relevant diseases started before Barocco randomization | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Relevant diseases started after Barocco randomization | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX | XX | xx | XX |
| Dermatological apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Visual apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Respiratory apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Cardiovascular apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Gastrointestinal apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Genitourinary apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Muscoloskeletal apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Endocrine apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Neurological apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Psychiatric apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Immunological apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Laboratory apparatus - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

# Statistical Analysis Plan BAROCCO

| | ARM A | ARM B | ARM C | Overall |
|----------------------------|-------|-------|-------|---------|
| Number of patients – n (%) | N=XX | N=XX | N=XX | N=XX |

**Legend:** ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects; SD: standard deviation. Q1 - Q3: First - third quartile. Min - Max: minimum - maximum values.

**Table 6. Tumour Characteristics – ITT Analysis Set** (table 14.1.2.2 CSR)

| CSR) | | | | |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
| Time from diagnosis (years) | | | | |
| Mean (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X<br>- XX.X) | XX.X (XX.X<br>- XX.X) | XX.X (XX.X<br>- XX.X) | XX.X (XX.X<br>- XX.X) |
| Min – max | XX.X-XX.X | XX.X-XX.X | XX.X-XX.X | XX.X-XX.X |
| Missing | xx | xx | xx | XX |
| Primary Site - n (%) | | | | |
| Ovary | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Fallopian | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Peritoneal | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | xx | xx | xx | xx |
| F.I.G.O. Stage - n (%) | | | | |
| IA | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IIA | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| AIII | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IB | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IIB | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IIIB | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IC | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IIC | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IIIC | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| IV | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | xx | xx | xx | xx |
| Missing | xx | xx | xx | xx |
| Histological Type - n (%) | | | | |
| Serous | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Endometroid | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mixed | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unspecified | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Mucinous | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Clear Cell | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Transitional | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unspecified | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Missing | XX | XX | XX | XX |

# Statistical Analysis Plan BAROCCO

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Size of residual disease after primary surgery - n (%) | | | | |
| <=1cm | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| >1cm | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | xx | xx | xx | xx |
| Missing | xx | xx | XX | XX |

**Legend:** ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects.
SD: standard deviation. Q1 - Q3: First - third quartile. Min - Max: minimum -

maximum values.
Table 7. Previous therapies – ITT Analysis Set (table 14.1.2.3 CSR) ARM B ARM C Overall ARM A N=XXN=XXN=XXN=XX **Previous** Chemotherapies lines n (%) Mean (SD) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX.X (XX.X XX.X (XX.X XX.X (XX.X -XXXX (XX.X Median (Q1 - Q3) - XX.X) - XX.X) - XX.X) XX.X) XX.X-XX.X XX.X-XX.X XX.X-XX.X XX.X-XX.X Min - Max Missing XX XX XX XX **Previous** Chemotherapies lines n (%) XX (XX.X) 2 XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) 3 XX (XX.X) 4 XX (XX.X) XX (XX.X) XX (XX.X) XX XXXXXX Missing Last line before Barocco - n (%) XX (XX.X) XX (XX.X) XX (XX.X) Monotherapy with PLATIN XX (XX.X) XX (XX.X) Associations with PLATIN XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX(XX,X)Monotherany without PLATIN XX (XX.X)

| | Monotnerapy without PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
|---|---|---|---|---|---|
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Previuos treatment<br>with antiangiogenic<br>drugs - n (%) | | | | |
| | No | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Yes | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Previuos chemotherapy<br>lines - n (%) | , | | | |
| | Three or more lines | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Up to 2 lines | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Line 1 | Number of patients - n<br>(%)<br>Previous Chemotherapi | XX (XX.X)<br>es - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Monotherapy with PLATIN Associations with | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | PLATIN Monotherapy without | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

| | Other | 10/ (0// 10 | 204 00000 | | |
|---|---|---|---|---|---|
| | | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | 101.001.0 | <b>101 00110</b> | | |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| Line 2 | Number of | 101.001.10 | 201 (2012) | | |
| | patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Previous Chemothera Monotherapy with | ipies - n (%) | | | |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Associations with | 70X (70X.X) | λλ (λλ.λ) | ^^ (^^.^) | ^^ (^^.^) |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Monotherapy without | | | | . , |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | ( | ( | 70. (70.07.) | 701 (70117t) |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Number of | | | | |
| Line 3 | | | | | |
| Line 3 | patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Line 3 | patients - n (%)<br>Previous Chemothera | ` , | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with | pies - n (%) | | , | |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN | ` , | XX (XX.X) XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with | xX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without | pies - n (%) | | , | |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN | xX (XX.X) | xx (xx.x) | XX (XX.X) | XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without | xx (xx.x)<br>xx (xx.x) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy | xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx (xx.x) xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx type - n (%) xx (xx.x) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| Line 3 | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx xx xx xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of patients - n (%) Previous Chemothera Monotherapy with | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of patients - n (%) Previous Chemothera Monotherapy with PLATIN | xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with PLATIN Monotherapy without PLATIN Other Missing Maintenance therapy Bevacizumab No Maintenance therapy Other Missing Number of patients - n (%) Previous Chemothera Monotherapy with PLATIN Associations with | xx (xx.x) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
|---|---|---|---|---|---|
| | Missing | XX | XX | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | , , | , , | | |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| Line 5 | Number of | | | | |
| Lille 3 | patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Previous Chemothera | pies - n (%) | | | |
| | Monotherapy with | | | VAL 401 VA | |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Associations with PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Monotherapy without | 777 (701.77) | 701 (701.71) | 701 (70171) | 701 (701.71) |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | хх | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | | | | |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| Line 6 | Number of | | | | |
| Line 0 | patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Previous Chemothera | pies - n (%) | | | |
| | Monotherapy with | VV (VV V) | VV (VV V) | VV (VV V) | VV (VV V) |
| | PLATIN Associations with | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Monotherapy without | , | , | ` , | , , |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | \0.40c++5 | \n, n, n, n | 10/ (20/ ) | \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |

| Line 7 | Number of patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
|---|---|---|---|---|---|
| | <b>Previous Chemothera</b> | pies - n (%) | ` , | , , | , , |
| | Monotherapy with | | | | |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Associations with | | | | |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Monotherapy without | | | | |
| | PLATIN | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |
| | Maintenance therapy | type - n (%) | | | |
| | Bevacizumab | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | No Maintenance | | ( , | | (/ |
| | therapy | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Other | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Missing | XX | XX | XX | XX |

Statistical Analysis Plan

Table 8. Previous therapies – Last Platinum free interval- ITT Analysis Set (table 14.1.2.4 CSR)

| ישחום סי בופאוסחה לוופוסחום בער בופרוותווו וויפט ווופו אמו די ו אוופול אום לוכחום די | | いんない しいの のうべき | こうしょうけん | _ |
|---|---|---|---|---|
| The second secon | ARM A | ARM B | ARM C | Overall |
| | N=XX | XX=N | N=XX | N=XX |
| Number of patients - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Last Platinum Free interval (months) | | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X-XX.X) | XX.X (XX.X-XX.X) | -X.X (XX.X-X-X-X-X-X-X-X-X-X-X-X-X-X-X-X-X-X- | XX.X (XX.X-XX.X) |
| Min – max | XXX - XXX | XX.X - XX.X | XXX - XXX | XXX - XXX |
| Missing | × | × | × | × |
| Time from last chemotherapy to first dose (months) | | | | |
| Mean (SD) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | - X.XX) X.XX<br>XX.X) | - XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X-XX.X | XXX-XXX | XX.X-XXX | XX.X-XXX |
| Missing | XX | XX | X | ×× |
| I amount ADM A. Daditavol. ADM B. Coditanih : Olaratin Continuous schodulo. ADM C. Coditanih Intermittent schodule. N. number of | | Tal diacaclo diacail | srmittent cchadul | o. M. nimbor of |

Table 9. Treatment Compliance - ITT Analysis Set (table 14.2.1.1 CSR)

| | | | | 1 1 |
|---|---|---|---|---|
| | AKM A | AKM B<br>N=XX | ARM C | Overall<br>N=XX |
| Never started - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | (x.xx) XX |
| Missing | ×× | × | × | × |
| Reasons: | | | | |
| Disease Progression | XX (xx.x) | XX (xx.x) | XX (xx.x) | (x.xx) XX |
| Adverse Event | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Intercurrent illness of sufficient severity | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Deterioration of clinical conditions | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Other Primary tumor occurrence | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Consent withdrawn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Patient refusal | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Lost at follow-up | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Death | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Other | × | × | × | × |
| Missing | XX | × | × | × |
| Treatment discontinued - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Missing | X | × | × | × |
| Reasons for discontínuation: | | | | |
| For ARM A – treatment completed | XX (xx.x) | | | |
| Disease Progression | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Adverse Event | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |

Statistical Analysis Plan BAROCCO

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Intercurrent illness of sufficient severity | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Deterioration of clinical conditions | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Other Primary tumor occurrence | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Consent withdrawn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Patient refusal | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Lost at follow-up | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Death | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Other | XX | × | × | × |
| Missing | X | × | × | X |
| Treatment completed - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Missing | X | ×× | × | × |
| Treatment ongoing - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Missing | X | XX | × | × |

Statistical Analysis Plan

Number of completed cycles in subjects who have discontinued the treatment – Compliance Analysis Set  $(table\ 14.2.1.2\ CSR)$ Table 10.

| X X X | | | |
|---|---|---|---|
| mber of patients - n (%) xxx (xxx) xxx (xxxx) mber of cycles xxx (xxxx) xxx (xxxxx) an (SD) xxx (xxxxx) xxx (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | ARM C | Overall |
| mber of patients - n (%) xxx (xxxx) mber of cycles xxx (xxxxx) an (SD) xxx (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | *************************************** | N=XX | N=XX |
| an (SD) X.X.X (XX.X.X.X.X.X.X.X.X.X.X.X.X.X.X.X. | | | |
| an (SD) X.X. (XX.X) dian (Q1 - Q3) X.X. X.X.X.X.X T - max mber of cycles - n (%) XX. X.X.X.X XX. X.X.X XX. X.X.X XX. XX.X XX. | | | |
| dian (Q1 - Q3) xx.x (xx.x-xx.x) xx.x-xx.x mber of cycles - n (%) xx (xx.x) | | XX.X (XX.X) | XX.X (XX.X) |
| mber of cycles - n (%) xx (xx.x) | XX.X (XX.X-XX.X) | XX.X (XX.X-XX.X) | XX.X (XX.X-XX.X) |
| mber of cycles - n (%) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | | XX.X-XX.X | XX.X-XX.X |
| XX (XXXX)<br>XX (XXXX)<br>XX (XXXX)<br>XX (XXXX)<br>XX (XXXXX) | | | |
| XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | | XX (XX.X) | XX (XX.X) |
| XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) | | XX (XX.X) | XX (XX.X) |
| XX (XX.X) XX (XX.X) XX (XX.X) | | XX (XX.X) | XX (XX.X) |
| XX (XX.X) XX (XX.X) | | XX (XX.X) | XX (XX.X) |
| XX (XX.X) | | XX (XX.X) | XX (XX.X) |
| | | XX (XX.X) | XX (XX.X) |
| | (X:XX) XX | XX (XX.X) | XX (XX.X) |
| (X:XX) XX | (XXXX) | XX (XX.X) | XX (XX.X) |
| (X.XX) XX | XX (XX.X) | xx (xxx.x) | xx (xx.x) |
| ≥10 XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

**Legend:** ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects; SD: standard deviation. Q1 - Q3: First - third quartile. Min - Max: minimum - maximum values.

Statistical Analysis Plan BAROCCO

Table 11. Dose intensity - Compliance Analysis Set (table 14.2.1.3 CSR)

| | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Number of patients - n (%) | a sussessing de melle de la constante de la co | | | |
| Paclitaxel | | | | |
| Mean (SD) | XX.X (XX.X) | | | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | | | XX.X (XX.X - XX.X) |
| Min – max | XX.X - XX.X | | | XXX - XXX |
| Missing | × | | | × |
| Cediranib | | | | |
| Mean (SD) | | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min – max | | XXX - XXX | XXX - XXX | X.X. i X.X |
| Missing | | × | × | × |

Statistical Analysis Plan BAROCCO

| | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | N=XX | XX = N | XX=N | N=XX |
| Olaparib | | | manuma ana a | — VARAN istandomum recens es es |
| Mean (SD) | | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min – max | | XX.X - XX.X | XX.X - XX.X | XXX - XXX |
| Missing | | × | × | × |

**Legend:** ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects; SD: standard deviation, Q1 - Q3: First - third quartile. Min - Max: minimum - maximum values.

Statistical Analysis Plan BAROCCO

XX (XX.X) XX (XX.X) XX (XX.X) (XXX) XX XX (XX.X) Overall X=X × XX (XX.X) (X.XX) XX (X.X) XX XX (XX.X) ARM C N=XX × Table 12. Progression Free Survival – ITT Analysis Set (table 14.2.2.1 CSR) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) (X.XX) XX XX (XX.X) XX (XX.X) (X.XX) XX XX (XX.X) XX (XX.X) XX (XX.X) XXII × XX (XX.X) (XXX) XX XX (XX.X) (XXX) XX XX (XX.X) XX (XX.X) XX (XX.X) ARM A XXIIN × Kaplan-Meier estimate of PFS (months) radiological progression for TL, NTL and NL radiological progression for NTL and NL radiological progression for TL and NTL Radiological progression for - n (%) radiological progression for TL and NL Progression or death - n (%) radiological progression for NTL radiological progression for TL radiological progression for NL Site of progression - n (%) no radiological progression Progression - n (%) Censored - n (%) Death - n (%) Multiple site Single site Missing

Statistical Analysis Plan

| The state of the s | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | XXIIN |
| 1st quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| Hazard ratio (Arm B vs. A) [95% CI] | | | | XX.X<br>[XX.X - XX.X] |
| P-value | | | | x.xxx |
| Hazard ratio (Arm C vs. A) [95% CI] | | | | XX.X<br>[XX.X - XX.X] |
| P-value | | | | X.XXX |

Statistical Analysis Plan BAROCCO

XX (XX.X) (XXX) XX Overall XII ×.× ××× × XX (XX.X) (X.XX) XX (XX.X) XX (XX.X) XXXXXXX (X.XX) XX XX (XX.X) XX (XX.X) (XXX) XX XX (XX.X) XX (XX.X) XX (XX.X) (XXXX) XX (XX.X) ARM C ×.× × × Table 13. Progression Free Survival - PP Analysis Set (table 14.2.2.2 CSR) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) (X.XX) XX (X.XX) XX XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) ARM B XXII ×.× ×.× × XX (XX.X) ARM A XXII X.X × × Kaplan-Meier estimate of PFS (months) radiological progression for TL, NTL and NL radiological progression for NTL and NL radiological progression for TL and NTL radiological progression for TL and NL Radiological progression for - n (%) Progression or death - n (%) radiological progression for NTL radiological progression for TL radiological progression for NL Site of progression - n (%) no radiological progression Progression - n (%) Censored - n (%) Death - n (%) 1st quartile Multiple site Median Single site Missing

Statistical Analysis Plan

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| Hazard ratio (Arm B vs. A) [95% CI] | | | | XXXX<br>XXXX |
| P-value | | | | xxx.x |
| Hazard ratio (Arm C vs. A) [95% CI] | | | | XX.X |
| P-value | | | | [v.vx - xxx.x |

Statistical Analysis Plan

Table 14. Progression Free Survival - Cox models - ITT Analysis Set (table 14.2.2.3 CSR)

| | a.c.pp. | Univariate | Univariate Analysis - PFS | | | Multivaria | Aultivariate Analysis - PFS | S: |
|---|---|---|---|---|---|---|---|---|
| | HR | 95% CI | X. | p-value | HR | 95% CI | CI | p-value |
| Covariate 1 | x.xx | xx.x | XX.X | x.xx | xx.x | xx.x | XX.X | x.xxx |
| Covariate 2 | xx.x | x:xx | xx.x | x.xxx | x.x | ××.× | XX.X | X.XXX |
| Covariate 3 | x.xx | xx.x | XX.X | x.xxx | XX.X | XX.X | XXX | x.xxx |
| Covariate n | X.X | XX.X | x:x | x.xx | xx.x | XX.X | XX.X | x.xxx |

Statistical Analysis Plan

Table 15. Progression Free Survival – Cox models - PP Analysis Set (table 14.2.2.4 CSR)

| | | Univaria | ariate Analysis - PFS | PFS Multivari | | Multivaria | Multivariate Analysis - PFS | PFS |
|---|---|---|---|---|---|---|---|---|
| | HR | 95 | 65% CI | p-value | H | 95% | 95% CI | p-value |
| Covariate 1 | xx.x | xx.x | X.XXX | x.xxx | XX.X | x.xx | XX.X | X.XXX |
| Covariate 2 | xx.x | ×.×. | x.xxx | x.xxx | x.x.x | x.x. | XX.X | x.xxx |
| Covariate 3 | x:xx | xx.x | x.xxx | x.xxx | xx.x | ×.× | XX.X | x.xx |
| Covariate n | xx.x | XX.X | x.xxx | x.xxx | ×.× | x:x | ××·× | x.xx |

Statistical Analysis Plan BAROCCO

Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects XX.X (XX.X) XX.X (XX.X) XX.X (XX.X) XX.X (xx.x) XXII ARM C XX.X (xx.x) XX.X (xx.x) XX.X (xx.x) XX.X (xx.x) ARM B (table 14.2.3.1 CSR) XX.X (XX.X) XX.X (XX.X) XX.X (XX.X) XX.X (xx.x) **ARM A** X=N Table 16. Response to treatment - ORR Analysis Set Response - n (%) SD

**Table 17. Objective response rate – ORR Analysis Set** (table 14.2.3.2 CSR)

| Response rate | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX | Chi-squared<br>Test |
|---|---|---|---|---|---|
| <b>CR+PR</b> - n (%) | XX.X (xx.x) | XX.X (xx.x) | XX.X (xx.x) | XX.X (xx.x) | Chi= xx.x |
| [95% CI] | [xx.x - xx.x] | [xx.x - xx.x] | [xx.x - xx.x] | | Df=xx |
| <b>SD + PD</b> - n (%) | XX.X (xx.x) | XX.X (xx.x) | XX.X (xx.x) | XX.X (xx.x) | P-value=<br>x.xxx |
| [95% CI] | [xx.x - xx.x] | [xx.x - xx.x] | [xx.x - xx.x] | | |

Table 18. Second Progression Free Survival – ITT Analysis Set (table

| 14.2.4.1 CSF | | | | |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
| Censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progression - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progression or death - n<br>(%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier estimate of PFS (months) | | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| Hazard ratio (Arm B<br>vs. A) [95% CI] | | | | XX.X<br>[XX.X -<br>XX.X] |
| P-value | | | | x.xxx |
| Harmad makin (Amar C | | | | XX.X |
| Hazard ratio (Arm C<br>vs. A) [95% CI] | | | | [XX.X -<br>XX.X] |
| P-value | | | | x.xxx |

**Table 19. Second Progression Free Survival – PP Analysis Set** (table 14.2.4.2 CSR)

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Censored - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progression - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Death - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Progression or death - n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Kaplan-Meier estimate of PFS (months) | | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| Hazard ratio (Arm B<br>vs. A) [95% CI] | | | | XX.X<br>[XX.X -<br>XX.X] |
| P-value | | | | x.xxx |
| Hazard ratio (Arm C | | | | XX.X |
| vs. A) [95% CI] | | | | [XX.X -<br>XX.X] |
| P-value | | | | x.xxx |

Statistical Analysis Plan BAROCCO

Table 20. Second Progression Free Survival - Cox models - ITT Analysis Set (table 14.2.4.3 CSR)

| | | Univariate | Jnivariate Analysis - PFS 2 | FS 2 | | Multivariat | Multivariate Analysis - PFS 2 | PFS 2 |
|---|---|---|---|---|---|---|---|---|
| | ¥ | 950 | 95% CI | p-value | HR | 95% | 95% CI | p-value |
| Covariate 1 | XXXX | xx.x | x.xx.x | x.xxx | XX.X | x.x. | XX.X | x.xxx |
| Covariate 2 | ×.× | x.x. | x.xxx | x.xxx | xx.x | xx.x | XX.X | x.xx |
| Covariate 3 | ×: XX | xx.x | x.xxx | x.xxx | ×:<br>×: | XX.X | XX.X | x.xxx |
| Covariate n | ×:× | ×.× | x.xxx | x.xxx | x.xx | ×.× | ×××× | x.xxx |

Statistical Analysis Plan BAROCCO

Table 21. Second Progression Free Survival - Cox models - PP Analysis Set (table 14.2.4.4 CSR)

| | | | אואמו ייי | Survival - COX IIIOUEIS - FF Allarysis SEL (Lable 14.2.4.4 CSK) | Notional And | שבר (ישחוב | 14.4.7.4 C. | 5K) |
|---|---|---|---|---|---|---|---|---|
| | | Univariate | Univariate Analysis - PFS 2 | FS 2 | | Multivariat | Multivariate Analysis - PFS 2 | PFS 2 |
| A CARLOS CONTRACTOR OF THE STATE OF THE STAT | HR | 950 | 95% CI | p-value | HR | 950 | 95% CI | p-value |
| Covariate 1 | x.xx | xx.x | X.XXX | x.xxx | XXX.X | xx.x | XX.X | x.xxx |
| Covariate 2 | XX.X | xx.x | X.XXX | X.XXX | X.XX | XX.X | XX.X | x.xx |
| Covariate 3 | x.xx | XX.X | X.XXX | x.xxx | XX.X | XX.X | XX.X | X.XXX |
| Covariate n | xx.x | xx.x | X.XXX | X.XXX | XXX. | x:xx | x.x | x.xxx |

Table 22. Overall Survival – ITT Analysis Set (table 14.2.5.1 CSR)

| | ARM A | ARM B | ARM C | Overal |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| Follow-up estimate<br>(months) | | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Censored - n (%) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X |
| Death - n (%) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X |
| Cause of death - n (%) | | | | |
| Disease- related | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Other | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Unknown | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Kaplan-Meier estimate of OS (months) | | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| · | | | | XX.X |
| Hazard ratio (Arm B vs.<br>A) [95% CI] | | | | [XX.X] |
| P-value | | | | x.xxx |
| ., , ,, ,, ,, | | | | XX.X |
| Hazard ratio (Arm C vs.<br>A) [95% CI] | | | | [XX.X<br>XX.X] |
| P-value | | | | x.xxx |

Table 23. Overall Survival – PP Analysis Set (table 14.2.5.2 CSR)

| | ARM A | ARM B | ARM C | Overall |
|---|---|---|---|---|
| | N=XX | N≃XX | N=XX | N=XX |
| Follow-up esti<br>(months) | mate | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Censored - n (%) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X |
| Death - n (%) | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX.X |
| Kaplan-Meier estimat<br>OS (months) | e of | | | |
| 1 <sup>st</sup> quartile | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X |
| 3 <sup>rd</sup> quartiles | XX.X | XX.X | XX.X | XX.X |
| Cause of death - n (%) | | | | |
| Disease- related | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Other | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Unknown | XX.X (XX.X) | XX.X (XX.X) | XX.X<br>(XX.X) | XX |
| Hazard ratio (Arm I | 2 .vo | | | XX.X |
| A) [95% CI] | ) vs. | | | [XX.X -<br>XX.X] |
| P-value | | | | x.xxx |
| Hazard ratio (Arm ( | · ve | | | XX.X |
| A) [95% CI] | . 43. | | | [XX.X -<br>XX.X] |
| P-value | | | | x.xxx |

Table 24. Overall Survival - Cox models - ITT Analysis Set (table 14.2.5.3 CSR)

| | | Univaria | Univariate Analysis - 0S | <b>S</b> 0 | | Multivaria | Multivariate Analysis - 0S | so - |
|---|---|---|---|---|---|---|---|---|
| | HR | 95% CI | o CI | p-value | HR | 95% CI | ° CI | p-value |
| Covariate 1 | XX.X | xx.x | xx.x | x.xxx | xx.x | ××.× | XX.X | x.xx |
| Covariate 2 | xx.x | XX.X | xx.x | x.xxx | xx.x | ××.× | XX.X | xxx.x |
| Covariate 3 | x.xx | xx.x | xx.x | x.xxx | XX.X | x.x | XX.X | x.xxx |
| Covariate n | xx.x | x.x | ××.× | x.xxx | ×.×. | ×.× | ××.× | x.xxx |

Statistical Analysis Plan

Table 25. Overall Survival - Cox models - PP Analysis Set (table 14.2.5.4 CSR)

| | *************************************** | Univaria | Univariate Analysis - 0S | SO | | Multivari | Multivariate Analysis - 0S | . os |
|---|---|---|---|---|---|---|---|---|
| orazione. | HR | 95% | 5% CI | p-value | HR | 95% | 95% CI | p-value |
| Covariate 1 | xx.x | xx.x | X'XX | x.xxx | XX,X | XX.X | XX.X | X.XXX |
| Covariate 2 | x.x. | x:xx | XX.X | x.xxx | xx.x | x.xx | XX.X | X.XXX |
| Covariate 3 | x.xx | xx.x | xx.x | XXXX | XX.X | xx.x | XX.X | X.XXX |
| Covariate n | XX.X | X'XX | XX.X | x.xxx | XX.X | XX.X | x.x | x.xx |

 $\overset{\circ}{\times}\overset{\circ}{\overset{\circ}{\times}}$ 

۳

×8×× 6××

×

×××

Statistical Analysis Plan BAROCCO

×.Χ ×.Χ . ×.Χ - X.X XX.X (X.X.X XX.X  $\overset{\times}{\times}\overset{\times}{\times}$ XX XX.X X Overail XX.X  $\overset{\times}{\times}\overset{\times}{\times}$ × × × ××× , ×× ×.× ×.× H × ×.× ×.× ×:× ×:×  $\overset{\times}{\times}\overset{\times}{\times}$  $\underset{\times}{\times}\underset{\times}{\times}\underset{\times}{\times}\underset{\times}{\times}$  $\stackrel{\text{\tiny $\times$}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}{\stackrel{\text{\tiny $\times$}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}{\stackrel{\text{\tiny $\times$}}}}}}}}}}}}}}}}}$  $\overset{\times}{\times}\overset{\times}{\times}$ XX.X ×× × , ×.×  $\overset{\times}{\times}\overset{\times}{\times}$ XXX  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ ×× ۳ × , XX.X XX.X  $\overset{\times}{\times}\overset{\times}{\times}$ ×.× ×.×  $\underset{\times}{\times}\underset{\times}{\times}\underset{\times}{\times}\underset{\times}{\times}$  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ , XX X.X 72 × ARM C X:XX X:XX ×:×× ×:×× ×8×× ×8×8  $\overset{\times}{\overset{\times}{\times}}\overset{\times}{\overset{\times}{\times}}$  $\overset{(x)}{\underset{(x,x)}{\times}}$ × × × ' XX.X) ×.× × 년 |-×××× ××× - X:XX  $\overset{\times}{\times}\overset{\widehat{\times}}{\times}$  $\overset{(x)}{\times}\overset{(x)}{\times}$ ××× × 10 Table 26. Quality of life - PRO Analysis Set (table 14.2.6.1 CSR) XXX  $\overset{\times}{\times}\overset{\times}{\times}$ ×.×.  $\times$  $\overset{(x)}{\times}\overset{(x)}{\times}$ (X:X ××× ××× ××× , XX XX.X Ë ×.× ×.×  $\overset{\times}{\times}\overset{\times}{\times}$  $\overset{\circ}{\times}\overset{\circ}{\times}$ XXX.X **T**2 × ARM B ×:× ×:× ×:× ×:× × × ×  $\overset{\times}{\times}\overset{\times}{\times}$ XX.X) X.X Ξ × X.X.X - X.X ×:×  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ (X:X ××× ××× 인 × , X.X.X , X.X.X  $\overset{(x)}{\times}\overset{(x)}{\times}$  $\times$  $\times$ ××× X:X × 23 (XXXX × (× × × × × × × ×.×. ×.×.  $\stackrel{\times}{\times}\stackrel{\times}{\times}$ ××× XX.X XX.X **T**2 × **ARM A** (X:XX X:XX X:XX ×.×. ×.×. ×.×. ×.×. ×.×. ×××, (X:X Ξ × - ×:× ×.×. ×.×. × (X X X X  $\overset{(x,x)}{\times}$ X:X  $\overset{\times}{\times}\overset{\times}{\times}$ X:X × 2 ţ (61 (01 ð Physical Well-being Mean (SD) Mean (SD) Min - Max Min - Max Median ( - Q3) Number patients Median - Q3) FACT-0 FACT-0 Missing (%) N 101

| Statistical Analysis Plan | BAROCCO |
|---------------------------|---------|
| | . –, |

| Missing xx xx xx | Social<br>Well-being | × (× × | XX.X XX.X XX.X Median (Q1 (XX.X (XX.X (XX.X - Q3) | XXX | Missing xx xx xx | Emotional<br>Well-being | | XX.X XX.X XX.X XX.X Median (Q1 (XX.X (XX.X (XX.X -Q3) Q3) | XXX |
|---|---|---|---|---|---|---|---|---|---|
| × | | | × | | × | | | ×× | |
| × | | ×××<br>××× | XXX | ××× | × | | ×××<br>×××<br>××× | X.X. , X. | XX.X<br>XX.X |
| × | | X.XX<br>X.XX | ××× | ` × | × | | XXXX<br>XXXX | ××× | XX.X<br>XX.X |
| × | | XX.X<br>(X.X.X | ×.×. , × | ××× | × | | × (× × | XXX, X | ××× |
| × | | ×:×<br>×:× | ×.×. , ×. | ××× | × | | ×.×.<br>×.×. | XXX , X | XX.X<br>XX.X |
| × | | XXXX<br>XXXX | XXX, X | XXX - X | × | | ×:XX | X.XX, , X | XX.X<br>XX.X |
| × | | ×××<br>××× | X.XX. , X | ××× | × | | × × × | × | ××× |
| × | | XXXX<br>XXXX | XXX. X | ××× | × | | ×:×<br>×:× | ×. × | XXX<br>XXX |
| × | | XXXX<br>XXXX | ××× × | X:X | × | | ×:XXX | XXX ' X | × |
| × | | × (× × | ××× , × | XX.X<br>XX.X | × | | ×:XXX | XXX , X | - X:XX |
| × | | × (× × | ××× , × | XXX | × | | ×.XXX | ×:×× | X X X |
| × | | ×××<br>×××<br>×××× | ×.×. ×. | XXXX<br>XXXX | × | | XXXX<br>XXXX | ××× | X:XX |
| × | | $\times \times $ | ××× | XXX | × | | ×××<br>××× | ××× , × | ×:× |

| Missing | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Functional<br>Well-being | | | | | | | | | | | | | | | | |
| Mean (SD) | × | × (× × | × (×<br>× | | ×.X.X | ×:×:<br>×:×: | ×××× | ×××<br>×××<br>×××× | ×.×.<br>×.×. | × (× × | ×.×.<br>×.×. | ×.×.<br>×.×. | ×××<br>××× | × | × × × | $\overset{\times}{\times}\overset{\times}{\times}$ |
| Median (Q1<br>- Q3) | × | ××× , | ×.×. , (x.×. | ×.×. (×.×. | ××× (××× , ×× | ×.×. , (x.×. ×. | ×.×. (x.×. | XXX, (XXX, XX, XX, XX, XX, XX, XX, XX, X | ×× | × | ××× (××× | ××× , (x<br>××× , (x | ×.×. (x.×. | ×.×. (x.×. | ××× (××× | × |
| Min - Max | ×:×<br>×:× | ×.×<br>×.× | ×:× | | XXX<br>XXX | XX.X<br>XX.X | XXX<br>XXX | XXXX<br>XXXX | XX.X<br>XX.X | ×.×. | ×××<br>××× | ×.×.<br>×.×. | ×××××××××××××××××××××××××××××××××××××× | ××××<br>×××× | XX.X<br>XX.X | XX.X<br>XX.X |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × | × |
| Ovarian<br>Cancer<br>Symptom<br>scales<br>Mean (SD)<br>Median (Q1<br>- Q3)<br>Min - Max<br>Missing | ×××× ×××× | ×(×,×, ×, | × ( | ×××× ××× × | × ( × | × ( × | × ( | × ( | ×××× , ××× × | × ( × | × | × ( | ×(\$\times\ti | ×××××××××××××××××××××××××××××××××××××× | × ( × × · ( × | ×××× × |
| Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib subjects | 1 A: Pacl | itaxel; Al | RM B: Ce | ediranib+ | Olaparib | | ous sche | Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of | IM C: Ce | diranib+( | Olaparib | Intermit | tent sche | edule; N | : number | of |

Statistical Analysis Plan BAROCCO

| FACT-0 | | ARM A | FACT-O ARM A ARM B ARM C | | ARM B | | | ARM C | | | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| es from<br>baseline<br>(T0) | T1-T0 | T2-T0 | T3-T0 | T1-T0 | 12-10 | T3-T0 | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 |
| Number<br>of<br>patients -<br>N (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (X:XX) | (xx.x) | XX (XX.X) | XX (xx.x) | XX (xx.x) XX (xx.x) XX (xx.x) | XX (xx.x) | × | × | × |
| Trial<br>Outcome<br>Index<br>(TOI) | | | | | | | | | | | | |
| Mean (SD) | ×.<br>×.<br>×.<br>×.<br>×. | ××× | ×.×.<br>×.×. | ×.×.<br>×.×. | × (× × | ××× | × | ×:XX<br>X:XX | ×:XX<br>XX:XX | ×.x.x | ×: X:<br>X: X: X: | ×.XX |
| Median<br>(Q1 - Q3) | ×:××<br>×:××<br>×:×× | XXXX<br>XXXX<br>XXXX | ×.×.<br>×.×.<br>×.×. | ×.×.×<br>×.×.×<br>×.×.× | ×.×.×<br>×.×.×<br>×.×.× | × | XX.XX<br>XX.XX | × | ×.×.×<br>×.×.×<br>×.×.× | × | ×.×.<br>×.×.× | × |
| Min - Max | XX.X - | XX.X<br>XX.X | | XX.X – | ×.×. | XX.XX | XX.X – | ×××<br>××× | XXX - XXX | ××× | ×.×. | ×.×. |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × |
| Physical<br>Well-<br>being | | | | | | | | | | | | |
| Mean (SD) | ×.×. | × (X × X | XXXX) | ×.×.<br>×.×. | × (× , × | ×.×.<br>(×.×. | ×××<br>(×××) | ×.X.X | ××× | × (× × | ×:XX | ×. (x. ×. ×. |

Statistical Analysis Plan BAROCCO

| FACT-0 | and the second s | ARM A | L. Carrier and T. Car | | ARM B | | | ARM C | | - Carlotte Control of the Control of | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| es from<br>baseline<br>(T0) | T1-T0 | T2-T0 | T3-T0 | T1-T0 | <b>T2-T0</b> | T3-T0 | T1-T0 | T2-T0 | 13-10 | T1-T0 | T2-T0 | T3-T0 |
| Median<br>(Q1 - Q3) | XX.X<br>- (XX.X<br>- (X.XX | XX.X<br>XX.X<br>XX.X | ×.×.<br>×.×.× | XX.X<br>(X.XX- | XXXX<br>XXXX<br>XXXX | XX.X<br>- XXXX | ×<br>×<br>×× | XX.X<br>(XX.X - | XX.X<br>(X.X. | - X:XX)<br>- X:XX) | XX.X<br>(X.XX<br>XX.X) | ×:×:<br>×:×:<br>×:×: |
| Min - Max | XX.X - | XX.X<br>XX.X | XX.X – | ××.×<br>××.× | XX.X<br>XX.X | ×.×. | XX.X<br>XX.X | XX.X<br>XX.X | ×.×. | ××××<br>×××× | ×××××××××××××××××××××××××××××××××××××× | ×:××<br>×:×× |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × |
| Social<br>Well-<br>being | | | | | | | | | | | | |
| Mean (SD) | ×.×. | ×.XX | ×.<br>×.<br>×.<br>×.<br>×.<br>×. | ×××× | ×.×.<br>×.×. | ×.X.X | ×.X.X | ×.X.<br>X.X. | XX.X<br>(X.XX) | ×:×:<br>×:×: | ×:XX<br>(X:XX) | XX.X<br>(X.X.X) |
| Median<br>(Q1 - Q3) | ×.×.<br>×.×.×<br>×.×.× | ×.×.<br>×.×.<br>×.×. | ××××<br>××××<br>×××× | ×:××<br>×:××<br>×:×× | ×.×.<br>×.×.×. | ×.×.<br>×.×.<br>×.×. | ××××<br>××××<br>×××× | ×××<br>×××<br>×××<br>××× | ×.×.<br>×.×.<br>×.×. | ×.×.×<br>×.×.× | × | ×:××<br>- (x:××<br>- x:×× |
| Min - Max | XX.X<br>XX.X | XX.X -<br>XX.X | XX.X<br>XX.X | XX.X<br>XX.X | ×.×. | ×××× | ×××× | ××××<br>×××× | ×:×<br>×:× | ×:×<br>×:× | XXX<br>XXX | ××<br>×× |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × |
| Emotiona<br>I | | | | | | | | | | | | |
| Well-<br>being | | | | | | | | | | | | |
| Mean (SD) | ××× | ×.×.<br>×.×. | ××××<br>×××× | ×.×.<br>(×.×. | ×.×.<br>×.×.× | ×:××<br>(×:××) | ×.×.<br>(×.×. | XX.XX<br>(XX.X) | ×:XX<br>X:XX | ×.×.<br>(×.×. | ×:××<br>(×:××) | ×:XX<br>X:XX |

Statistical Analysis Plan BAROCCO

| FACT-0<br>differenc | | ARM A | | | ARM B | | | ARM C | | | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| es from<br>baseline<br>(T0) | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 |
| Median<br>(Q1 - Q3) | XX.X<br>(X.X.X. | XX.X<br>(X.X.X<br>XX.X) | XX.X<br>(X.XX - X.X) | XX.X<br>(XX.X - | XXXX<br>XXXX-<br>XXXX | XX.X<br>(XX.X<br>- XXX) | XX.XX<br>XX.XX | XX.X<br>- (X.XX | - (X:XX)<br>- (X:XX) | XXXX<br>- (X:XX | × | XX.XX<br>XX.XX |
| Min - Max | ××<br>×× | XX.X – | ××<br>×× | ×.×.× | - ×:××<br>×:×× | ×××× | XX.X – | ×××× | - ×:××<br>×:×× | ×.×. | ×.×. | ×.×. |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × |
| Functiona<br>I<br>Well-<br>being | | | | | | | | | | | | |
| Mean (SD) | ×:×× | ×××<br>××× | ××× | ×.XX | ×××<br>×××<br>××× | ××× | ×.×. | ×.×.×. | XXXX<br>XXXX | × (X<br>XXXX | ×.XX<br>X.XX | ×:XX<br>X:XX |
| Median<br>(Q1 - Q3) | XX.X<br>XX.X<br>XX.X) | ××××<br>××××<br>×××× | ×:××<br>×:××<br>×:×× | ×.×.<br>×.×.× | ×.×.×<br>×.×.×<br>×.×.× | ×.×.<br>×.×.× | XX.X<br>XX.X<br>- XX.X | ×<br>××<br>×× | ××××<br>××××<br>×××× | × | × | × |
| Min - Max | ×.×. | ××<br>×.×× | ××<br>×.×× | ×××× | ×.×. | XX.XX<br>XX.X | - X.X.X<br>- X.X.X | XX.XX | XX.X<br>XX.X | - ×:<br>×:<br>×:<br>×: | ×××× | ×.×. |
| Missing | × | × | × | × | × | × | × | × | × | × | × | × |
| Ovarian<br>Cancer<br>Symptom<br>scales | | | | | | | | | | | | |

Statistical Analysis Plan BAROCCO

| FACT-0 | A A LIBERT A LIVE OF THE LIVE | ARM A | | | ARM B | | | ARM C | | | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| es from<br>baseline<br>(T0) | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 | T1-T0 | T2-T0 | T3-T0 |
| Mean (SD) | XXXX) | XX.X) | XXXX<br>(XXXX) | x:xx<br>(x:xx) | ×.XX | XX.X) | XX.X) | XX.X<br>(XX.X) | ×.<br>×.<br>×.<br>×. | ×.<br>×.<br>×.<br>×. | ×.×.×<br>×.×.× | ×:×<br>×:×<br>×:× |
| Median<br>(Q1 - Q3) | ×.×.×<br>×.×.×<br>×.×.× | ×.×.<br>×.×.×<br>×.×.× | ×.×.×<br>×.×.×<br>×.×.× | ×<br>×<br>× | ×.×.×<br>×.×.×<br>×.×.× | ×.×.<br>×.×.<br>×.×. | ×.×.<br>×.×.<br>×.×. | ×:××<br>×:××<br>×:×× | ×.×.×<br>×.×.×<br>×.×.× | ×.×.×<br>×.×.×<br>×.×.× | ×.×.×<br>×.×.×<br>×.×.× | ×:×:<br>×:×:× |
| Min - Max | ×.×.<br>×.×. | XX.X - | XX.X<br>XX.X | ××<br>×× | ×.×. | ×.×<br>×.× | ×××× | ×:×<br>×:× | ×:×<br>×:× | ×××××××××××××××××××××××××××××××××××××× | ×:.×<br>×:.× | ××<br>×× |
| Missing | × | × | × | × | X | × | × | × | XX | X | X | X |

Legend: ARM A: Paclitaxel, ARM B: Cediranib+Olaparib Continuous schedule, ARM C: Cediranib+Olaparib Intermittent schedule, N: number of s ubjects,SD: stadard deviation, Q1-Q3: First -third quartile, Min-Max: minimum - maximum values, T0: Time 0 (Baseline), T1: after 4 weeks, T2: after 8 weeks, T3: after 12 weeks.

Statistical Analysis Plan

Table 28. Quality of life - Mixed model for differences from baseline - PRO Analysis Set (table 14.2.6.3 CSR)

| ו מחום לסי לחשוונא מו ווופ " ואוצפת וווסמפו וכ | I or differences from baseline - PRO Analysis set (table 14.2.6.3 CSK) | PRO Analysis set (table | 14.7.5.3 CSK) |
|---|---|---|---|
| FACT-O scores | Effect | Estimate [95% CI] | P-value |
| | Intercept | XX [XX.XX-XX-XX] | X.XXX |
| Trial outcome index (TOT) | Treatment | xx [xx.xx-xx-xx] | X.XX |
| | Time | XX [XX.XX-XX-XX] | X.XX |
| | Interation | XX [XX.XX-XX-XX] | X,XXX |
| | Intercept | XX [XX.XX-XX-XX] | x.xx |
| Dhysical Well-being | Treatment | XX [XX.XX-XX-XX] | X.XXX |
| | Time | XX [XX.XX-XX-XX] | X.XXX |
| | Interation | XX [XX.XX-XX-XX] | X.XXX |
| | Intercept | XX [XX:XX-XX-XX] | X,XXX |
| Social Well-heing | Treatment | XX [XX.XX-XX-XX] | x.xxx |
| | Time | XX [XX.XX-XX-XX] | X.XXX |
| | Interation | XX [XX.XX-XX-XX] | X.XXX |
| | Intercept | XX [XX.XX-XX-XX] | x.xxx |
| Emotional Well-haind | Treatment | XX [XX.XX-XX-XX] | X.XXX |
| | Time | XX [XX.XX-XX-XX] | X.XXX |
| | Interation | XX [XX.XX-XX-XX] | X.XXX |
| | Intercept | XX [XX.XX-XX-XX] | X.XXX |
| Finctional Well-baing | Treatment | XX [XX.XX-XX-XX] | X.XXX |
| | Time | XX [XX:XX-XX-XX] | x.xxx |
| | Interation | XX [XX.XX-XX-XX] | x.xxx |
| | Intercept | XX [XX.XX-XX-XX] | X.XXX |
| Ovarian Cancer Symptom scales | Treatment | XX [XX.XX-XX-XX] | x.xxx |
| | Time | XX [XX.XX-XX-XX] | X.XXX |
| | Interation | XX [XX.XX-XX] | x.xxx |
| Legend: ARM A: Paclitaxel, ARM B: Cediranib+Olaparib Continuous schedule, ARM C: Cediranib+Olaparib Intermittent schedule, N: number of | ib Continuous schedule, ARM C: Cedira | inib+Olaparib Intermittent sche | dule, N: number of |
| 100,000 | | | |

subjects.

Statistical Analysis Plan

Table 29. Number of evacuations per day - Safety 1 Analysis Set (table 14.3.1.1 CSR)

| | a May | CMGV | OVERALI |
|---|---|---|---|
| | Z = N | N=8 | N=15 |
| Number of daily stools at baseline | | | |
| | (X:XX) XX | (XXXX) XX | XX (XX.X) |
| Missing | × | × | × |
| Total number of evacuations | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XXX - XXX | XXX - XXX |
| Missing | × | × | × |
| Total number of evacuations in cycle 1 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | (X.X X.X.) XXX (XX.X - XX.X) XXX (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Mín - Max | XXX - XXX | XX.X - XX.X | XXX - XXX |
| Missing | ×× | × | ×× |
| Total number of evacuations in cycle 2 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XXX - XXX | XX.X - XX.X | XX.X - XX.X |
| Missing | × | × | X |
| Total number of evacuations in cycle 3 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |

Statistical Analysis Plan BAROCCO

| | ARM B<br>N=7 | ARM C<br>N=8 | OVERALL<br>N=15 |
|---|---|---|---|
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| Missing | × | × | × |
| Total number of evacuations in cycle 4 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XXX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XXX - XXX | XX.X - XX.X |
| Missing | × | × | × |
| Total number of evacuations in cycle 5 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XXX - XXX | XX.X - XX.X |
| Missing | × | × | × |
| Total number of evacuations in cycle 6 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| Missing | × | × | × |
| Total number of evacuations in cycle 7 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
Statistical Analysis Plan BAROCCO

| | ARM B<br>N=7 | ARM C<br>N=8 | OVERALL<br>N=15 |
|---|---|---|---|
| Min - Max | XXX - XXX | XXX - XXX | XX.X - XX.X |
| Missing | X | × | × |
| Total number of evacuations in cycle 8 | | | |
| Mean (SD) | XXX (XXX) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XXX - XXX | XXX - XXX |
| Missing | × | × | × |
| Total number of evacuations in cycle 9 | | | |
| Mean (SD) | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | (X.X XX.X) X.XX | XX.X (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XX.X - XX.X | XXX - XXX | XXX - XXX |
| Missing | X | × | × |
| Total number of evacuations in cycle 10 | | | |
| Mean (SD) | XXX (XXX) | XX.X (XX.X) | XX.X (XX.X) |
| Median (Q1 - Q3) | XXX - XXXX | (X.XX - XX.X) XXX (XX.X - XX.X) XXX (XX.X - XX.X) | XX.X (XX.X - XX.X) |
| Min - Max | XXX - XXX | XX.X - XX.X | XXX - XXX |
| Missing | × | × | × |
| Worst experienced grade of diarrhea according to NCI-CTCAE | | | |
| 0 | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| | XX.X (XX.X) | XX.X (XX.X) | XX.X (XX.X) |
| 2 | XXX (XXX) | XX.X (XX.X) | XX.X (XX.X) |

Statistical Analysis Plan BAROCCO

| | ARM B<br>N=7 | ARM C<br>N=8 | OVERALL<br>N=15 |
|---|---|---|---|
| ಣ | XX.X (XX.X) | (X:XX) X:XX | (X.XX) X.XX |
| Missing | × | × | × |
| Legend: ARM B: Cediranib+Olaparib Continuous schedule, ARM C: Cediranib+Olaparib Intermittent schedule, N: number of subjects, SD: stadard deviation, Q1-Q3: First -third quartile, Min-Max: minimum - maximum values. | ım - maximum values | | |

Statistical Analysis Plan BAROCCO

Table 30. Change of evacuations per day - Safety 1 Analysis Set (table 14.3.1.2 CSR)

| Number of evacuations per day | ARM B<br>N=XX | ARM C<br>N=XX | T-test<br>p-value |
|---|---|---|---|
| Score | Mean (SD) | Mean (SD) | |
| Number of evacuations per day | XX (xx.x) | (x·xx) XX | x.xxx |
| Legend: ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: total number of subjects | ittent schedule; N: | total number of s | ubjects |

Statistical Analysis Plan BAROCCO

Table 31, Adverse reactions - Safety 2 Analysis Set (table 14.3.1.3 CSR)

| | | <b>G1</b> | 62 | 63 | <b>G</b> 4 | G3+G4 | Chi-squared |
|---|---|---|---|---|---|---|---|
| | Atin | n (%) | u (%) | n (%) | n (%) | (%) u | for trend |
| OVERALL | ARM A | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | x.xxx |
| | ARM B | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| en area de la desta de de Candidatel Incolares de anticidades de la composition della composition dell | ARM C | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| SOC1 | ARM A | (xx) xx | (x) xx | (x) xx | (x) x | (x) xx | <b>X.XXX</b> |
| | ARM B | (xx) xx | ( <del>x</del> ) <del>x</del> | (x) x | (x) xx | (x) x | |
| | ARM C | ( <del>xx</del> ) <del>xx</del> | (xx) xx | (xx) xx | ( <del>x</del> ) x | (x) xx | |
| PREFERRED TERM1 | ARM A | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | xxxx |
| | ARM B | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| | ARM C | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| PREFERRED TERM2 | ARM A | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (x) x | ××× |
| | ARM B | ( <u>x</u> ) x | (xx) xx | (xx) xx | (x) x | ( <del>x</del> ) xx | |
| | ARM C | (xx) xx | (xx) xx | (xx) xx | (x) xx | (xx) xx | |
| PREFERRED TERMn | ARM A | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | x.xxx |
| | ARM B | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| | ARM C | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| Socn | ARM A | ( <u>x</u> ) x | ( <u>xx</u> ) <u>xx</u> | ( <del>x</del> ) <del>xx</del> | (xx) xx | (xx) xx | XXX |
| | ARM B | ( <del>xx)</del> <del>xx</del> | ( <u>X</u> X | ( <u>x</u> ) xx | (x) xx | (xx) xx | |
| | ARM C | ( <b>※</b> ) <b>※</b> | (x) xx | ( <u>x</u> ) x | (xx) xx | (xx) xx | |
| PREFERRED TERMn | ARM A | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | ×××× |

Statistical Analysis Plan BAROCCO

| **** | <b>G1</b> | <b>G2</b> | 63 | <b>Q</b> | 63+64 | Chi-squared |
|-------|-----------|-----------|---------|----------|---------|-------------|
| E C | n (%) | n (%) | (%) п | (%) u | (%) u | for trend |
| ARM B | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |
| ARM C | (xx) xx | (xx) xx | (xx) xx | (xx) xx | (xx) xx | |

**Legend**: ARM A: Paclitaxel, ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: total number of subjects

Statistical Analysis Plan

Table 32. Overview of Serious Adverse Events - Safety 2 Analysis Set (table 14.3.1.4 CSR)

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Number of patients - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SAEs - n | × | × | × | × |
| Subjects with at least one SAE - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SADRs - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SUSARs - n (%) | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| <b>Legend</b> : ARM A: Paclitaxel, ARM B: Cediranib+Olaparib Continuous sof subjects | parib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: total number | b+Olaparib Intermitt | ent schedule; N: t | otal number |

Statistical Analysis Plan BAROCCO

Table 33. Description of Serious Adverse Events (SAEs) - Safety 2 Analysis Set (table 14.3.1.5 CSR)

| lable 33. Description of Serious Auverse Evelits (SAES) - Safety 2 Analysis Set (Abbe 14:0:1:0 CM) | (SAES) - Saicily & | שומאוסודע | נמטוט דידיטיים מטמט | N |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
| Causal relationship - n (%) | | | | |
| With only disease | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| With only Paclitaxel | XX (xx.x) | | | XX (xx.x) |
| With both disease and Paclitaxel | XX (xx.x) | | | XX (xx.x) |
| With only Olaparib | | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| With both disease and Olaparib | | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| With only Cediranib | | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| With both disease and Cediranib | | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| With disease, Olaparib and Cediranib | | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Seriousness - n (%) | | | | |
| Death | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Hospitalisation/Prolonged hospitalisation | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |

Statistical Analysis Plan BAROCCO

| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
|---|---|---|---|---|
| Life-threatening | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Medically Significant | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Significant disability | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Congenital anomaly/birth defect | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Death | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continusubjects | varib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of | ediranib+Olaparib Inter | rmittent schedule; N | l: number of |

Statistical Analysis Plan BAROCCO

Table 34. Description of Serious Adverse Events (SAEs) by MedDRA – Safety 2 Analysis Set (table 14.3.1.6

| CSK) | | | **** | |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall<br>N=XX |
| SAEs by MEdDra System Organ Class (SOC) - n (%) | | | | |
| SOC1 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SOC2 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SOCn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SAEs by MEdDra Preferred Term (PT) - n (%) | | | | |
| PT1 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| PT2 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| PTn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of | inuous schedule; ARM C | Cediranib+Olaparib Int | rermittent schedule; | N: number of |

subjects

| Table 35. Description of Serious Adverse Drug $CSR$ | Reactions (SADRs) - Safety 2 Analysis Set (table 14.3.1.7 | s) - Safety 2 An | alysis Set $(\it tal$ | ble 14.3.1.7 |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C | Overall<br>N=XX |
| NCI/CTC grade - n (%) | | | · A management of the state of | And the second s |
| 1 – Mild | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| 2 - Moderate | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| 3 – Severe | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| 4 - Life-treatening | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| 5 - Fatal | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Outcome - n (%) | | | | |
| Resolved | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Resol. With sequelae | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Not resolved | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Fatal | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| Unknown | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |

Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects

Statistical Analysis Plan

Table 36. Description of Serious Adverse Drug Reactions (SADRs) by MEdDra – Safety 2 Analysis Set (table 14.3.1.8 CSR)

| 14.3.1.8 CSK) | | | | |
|---|---|---|---|---|
| | ARM A<br>N=XX | ARM B<br>N=XX | ARM C<br>N=XX | Overall N=XX |
| SADRs (Serious Adverse Drug Reactions) - n (%) | ×× | X | X | × |
| SADRs by MEdDra System Organ Class (SOC) - n (%) | | | | |
| SOC1 | (x.xx) XX | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SOC2 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SOCn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| SAERs by MEdDra Preferred Term (PT) - n (%) | | | | |
| PT1 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| PT2 | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| PTn | XX (xx.x) | XX (xx.x) | XX (xx.x) | XX (xx.x) |
| | | The second communication and the second seco | ASSESSMENT OF THE PROPERTY OF | ************************************** |

Legend: ARM A: Paclitaxel; ARM B: Cediranib+Olaparib Continuous schedule; ARM C: Cediranib+Olaparib Intermittent schedule; N: number of subjects

## 7. APPENDIX B: LISTINGS OF SECTION 16.2 OF THE CSR

Overall content of Appendix 16.2 of the CSR (see guideline ICH topic E3):

- 16.2.1 Discontinued patients
- 16.2.2 Protocol Deviations
- 16.2.3 Patients Excluded from the Efficacy Analysis
- 16.2.4 Demographic Data / Tumor characteristics
- 16.2.5 Compliance
- 16.2.6 Individual Efficacy Response Data
- 16.2.7 Adverse Events Listings (each patient)

| Listing<br>Number | Listing Title | Section<br>of the<br>CSR | Page |
|---|---|---|---|
| _ | Subject disposition (All subjects set) | 16.2.1 | 87 |
| | . Protocol Deviations | 16.2.2 | 88 |
| | Inclusion criteria (All subjects set) | 16.2.2 | 89 |
| Listing 4 | Exclusion criteria (All subjects set) | 16.2.2 | 90 |
| Listing 5 | Patients inclusion in the analysis sets (All subjects set) | 16.2.3 | 91 |
| Listing 6 | Demographic and baseline characteristics (All subjects set) | 16.2.4 | 92 |
| Listing 7 | Tumor characteristics (All subjects set) | 16.2.4 | 93 |
| | Previous therapies (All subjects set) | 16.2.4 | 94 |
| Listing 9 | Drug administration: dose administer per cycle (All subjects set) | 16.2.5 | 95 |
| Listing<br>10 | Treatment compliance (All subjects set) | 16.2.5 | 96 |
| Listing<br>11 | Efficacy data (All subjects set) | 16.2.6 | 97 |
| Listing<br>12 | Follow-up (All subjects set) | 16.2.6 | 98 |
| Listing<br>13 | Response to treatment (All subjects set) | 16.2.6 | 99 |
| Listing<br>14 | Tumor assessment (All subjects set) | 16.2.6 | 100 |
| Listing<br>15 | Quality of life assessment: FACT-O scores (All subjects set) | 16.2.6 | 101 |
| Listing<br>16 | Quality of life assessment: FACT-O items (All subjects set) | 16.2.6 | 102 |
| Listing<br>17 | Number of evacuation per day (All subjects set) | 16.2.7 | 103 |

| Listing<br>Numbe | r Listing Title | Section of the CSR | Page |
|---|---|---|---|
| Listing<br>18 | Treatment tolerability- haematological toxicity (All subjects set) | 16.2.7 | 104 |
| Listing<br>19 | Treatment tolerability- Non haematological toxicity (All subjects set) | 16.2.7 | 105 |
| Listing<br>20 | Serious Adverse Events | 16.2.7 | 106 |

Statistical Analysis Plan BAROCCO

Listing 1. Subject disposition (All subjects set) (listing 16.2.1.1)

| Lost to Fup | Information of the Annual Construction of the Constitution of the |
|---|---|
| N Fup | Second the second secon |
| N cycles | |
| Reason for<br>withdrawal | |
| Status | |
| Arm | |
| Age | Approximately and the second s |
| Key | |

Statistical Analysis Plan

Statistical Aliatysis Fri BAROCCO

Listing 2. Protocol Deviations (listing 16.2.2.1)

| Deviation: specification | The state of the s |
|---|---|
| Deviation | |
| Arm | |
| Age | amma ayama enganyayayayayayayayayayayayayayayayayaya |
| Key | |

Statistical Analysis Plan BAROCCO

Listing 3. Inclusion criteria (All subjects set) (listing 16.2.2.2)

| | Inclusion n<br>(yes/no) |
|---|-------------------------|
| | Inclusion 6<br>(yes/no) |
| | Inclusion 5<br>(yes/no) |
| | Inclusion 4<br>(yes/no) |
| | Inclusion 3<br>(yes/no) |
| | Inclusion 2<br>(yes/no) |
| | Inclusion 1<br>(yes/no) |
| | Arm |
| | Age |
| 1 | Key |

Statistical Analysis Plan

Listing 4. Exclusion criteria (All subjects set) (listing 16.2.2.3)

| į | ()<br>() | V. | Exclusion 1 | Exclusion 2 | Exclusion 3 | Exclusion 4 | Exclusion 5 | Exclusion 6 | Exclusion n |
|---|---|---|---|---|---|---|---|---|---|
| ,<br>u | ⊒ñ€ | Ę | (yes/no) | (yes/no) | (yes/no) | (yes/no) | (yes/no) | (yes/no) | (yes/no) |

Statistical Analysis Plan BAROCCO

Listing 5. Patients inclusion in the analysis sets (All subjects set) (listing 16.2.3.1)

| 1 | | | | | *************************************** | | ì | | |
|---|---|---|---|---|---|---|---|---|---|
| 2 | ( ) | 4 e | All subjects<br>analysis set | Intent-to-treat<br>analysis set | Per-protocol<br>analysis set | Safety analysis<br>set | Overall Response rate analysis set | Compliance<br>analysis set | PRO analysis<br>set |
| Á<br>e<br>v | D<br>O | <u> </u> | yes/no/if no<br>reason) | (yes/no/if no<br>reason) | (yes/no/if no<br>reason) | (yes/no/if no<br>reason) | (yes/no/if no<br>reason) | (yes/no/if no<br>reason) | (yes/no/if no<br>reason) |

Listing 6. Demographic and baseline characteristics (All subjects set) (listing 16.2.4.1)

Dataset Characteristic n Characteristic1 Arm Age Key

Statistical Analysis Plan BAROCCO

Listing 7. Tumor characteristics (All subjects set) (listing 16.2.4.2)

| Dataset |
|------------------|
| Characteristic n |
| Characteristic1 |
| Arm |
| Age |
| Key |

Statistical Analysis Plan

Listing 8. Previous therapies (All subjects set) (listing 16.2.4.3)

| Dataset | |
|---|---|
| Therapy n | WANTERSON TO THE WASTE OF THE W |
| Therapy 1 | |
| Arm | |
| Age | out til til se en |
| Key | |

Statistical Analysis Plan BAROCCO

Listi

| | Dataset |
|---|---|
| 6,2,5,1) | Treatment not administered |
| .) (listing 1 | Dose<br>modification |
| dose administer per cycle (All subjects set) (listing 16.2.5.1) | Time<br>modification |
| er cycle (All | Treatment<br>modification<br>(yes/no) |
| nister p | Dose<br>Olaparib |
| dose admir | Dose<br>Cediranib |
| ration: ( | Dose<br>Paclitaxel |
| ıdminist | Date |
| Drug a | Arm |
| ing 9. | Age |
| List | Key |

Statistical Analysis Plan

| | Dataset |
|---|---|
| | Dose<br>Intensity<br>Olaparib |
| | Dose<br>Intensity<br>Cediranib |
| 2.5.2) | Dose<br>Intensity<br>Paclitaxel |
| iance (All subjects set) (listing 16.2.5.2) | Reason for<br>modification |
| cts set) ( | N cycles |
| (All subje | Treatment<br>modification |
| | Treatment |
| Listing 10. Treatment compl | Arm |
| 10. Trea | Age |
| Listing | Key |

Statistical Analysis Plan BAROCCO

Listing 11. Efficacy data (All subjects set) (listing 16.2.6.1)

| Dataset |
|-----------------------------------------------|
| Progression free<br>survival<br>time (months) |
| Date of<br>progression |
| Progression |
| Cause of<br>death |
| Overall<br>survival time<br>(months) |
| Date of<br>death |
| Death De |
| Arm |
| Age |
| Key |

Statistical Analysis Plan

Listing 12. Follow-up (All subjects set) (listing 16.2.6.2)

| Dataset | |
|---|---|
| Second<br>Progression free<br>survival<br>time (months) | |
| Date of second<br>progression | |
| Second<br>Progression | |
| Cause of<br>death | |
| Overall survival time (months) | |
| Date of<br>death | |
| Death | THE RESERVE THE PROPERTY OF THE PERSON NAMED IN THE PERSON NAMED I |
| Arm | |
| Age | |
| Key | |

Statistical Analysis Plan BAROCCO

Listing 13. Response to treatment (All subjects set) (listing 16.2.6.3)

| Dataset |
|------------------------------------|
| Event (progression/death/censored) |
| Response<br>duration<br>(months) |
| Reason for no<br>response |
| Best response |
| Arm |
| Age |
| Key |

Statistical Analysis Plan

Listing 14. Tumor assessment (All subjects set) (listing 16.2.6.4)

| Dataset |
|----------------------------------------|
| Overall evaluation |
| Conclusion for<br>new lesion |
| Conclusion for<br>non-target<br>lesion |
| Conclusion for target lesion |
| date |
| Evaluation<br>(weeks) |
| Arm |
| Age |
| Key |

Statistical Analysis Plan BAROCCO

Listing 15. Quality of life assessment: FACT-O scores (All subjects set) (listing 16.2.6.5)

| | Dataset |
|----|--------------------------|
| | Additional concern |
| | Emotional well-<br>being |
| | Functional<br>well-being |
| | Social well-<br>being |
| | Physical<br>well-being |
| | TOI |
| | date |
| | Evaluation<br>(weeks) |
| | Arm |
| | Age |
| ,, | Key |

Statistical Analysis Plan

| _ |
|---------------------------------------|
| 2.6.6) |
| 9 |
| N |
| 16 |
| ₫ |
| Ξ |
| <u>S</u> |
| t) (listi |
| £ |
| s set |
| Ŋ |
| Ü |
| 5 |
| 3 |
| <b>5</b> |
| S II S |
| <u>'</u> |
| Ε |
| te |
| <u>.</u> |
| U |
| ment: FACT-C |
| ment: FACT-C |
| ment: FACT-C |
| assessment: FACT-C |
| ment: FACT-C |
| assessment: FACT-C |
| assessment: FACT-C |
| assessment: FACT-C |
| assessment: FACT-C |
| uality of life assessment: FACT-C |
| lity of life assessment: FACT-C |
| 6. Quality of life assessment: FACT-C |
| . Quality of life assessment: FACT-C |
| 6. Quality of life assessment: FACT-C |
| 6. Quality of life assessment: FACT-C |

| | Dataset |
|---|---|
| 2.6.6) | Item 39 |
| (listing 16 | Item |
| isessment: FACT-O items (All subjects set) (listing 16.2.6.6 | Item 3 |
| ms (All su | Item 2 |
| FACT-0 ite | Item 1 |
| sment: | date |
| life assess | Evaluation<br>(weeks) |
| ality of life as | Arm |
| 16. Qu | Age |
| isting | Key |

Statistical Analysis Plan BAROCCO

Listing 17. Number of evacuation per day (All subjects set) (listing 16.2.7.1)

| Dataset |
|-----------------------------------|
| Worst grade<br>(NCI-CTCAE) |
| Number of days<br>of Loperamid |
| Dose<br>Loperamid |
| Number of<br>days |
| Total number<br>of<br>evacuations |
| date |
| Evaluation<br>(weeks) |
| Arm |
| Age |
| Key |

Statistical Analysis Plan

Statistical Analysis I BAROCCO

Listing 18. Treatment tolerability- haematological toxicity (All subjects set) (listing 16.2.7.2)

| Toxicity n |
|------------|
| Toxicity 1 |
| Arm |
| Age |
| Key |

Dataset

Statistical Analysis Plan

Listing 19. Treatment tolerability- Non haematological toxicity (All subjects set) (listing 16.2.7.3)

| Dataset |
|------------|
| Toxicity n |
| Toxicity 1 |
| Arm |
| Age |
| Key |

Statistical Analysis Plan BAROCCO

Listing 20. Serious Adverse Events (listing 16.2.7.4)

| Outcome |
|-------------------|
| Severity Outcome |
| Seriousness |
| tion Relationship |
| Description |
| Arm |
| Age |
| Key |

## 8. APPENDIX C: FIGURES TEMPLATE

Figure 2. Kaplan-Meier display of Progression Free Survival – <u>ITT</u> Analysis Set



Figure 3. Kaplan-Meier display of Progression Free Survival –  $\underline{PP}$  Analysis Set



Figure 4. Kaplan-Meier display of Second Progression Free Survival – <u>ITT</u> Analysis Set



Figure 5. Kaplan-Meier display of Second Progression Free Survival  $-\underline{PP}$  Analysis Set







